## Researchers:

# Eliseth Ribeiro Leão Lidiane Soares Sodré da Costa

Evidence-Based Practice: Proposed Application of Facilitating Tools for Clinical Nurses

Plataforma Brasil - Approval Number: 26787019.5.0000.0071

Board Affiliation: Research Ethics Committee of Hospital Israelita Albert Einstein

## 1. INTRODUCTION

The adoption of Evidence-Based Practice (EBP) is widely used to improve the quality and safety of health care, including the reduction of avoidable costs. (1)

A PBE has its origins in medicine used in tests and has been defined as "the conscientious and judicious use of the best discoveries made in decision-making in the individual care of patients". (1, 2)

Despite the fact that hospitals are considered responsible for delivering the best services available in the health area and based on use, signs of only a small percentage of health professionals are consistently doing this. (1, 2)

Many barriers are encountered in real practice, including time constraints, lack of personal motivation, professional resistance to research and knowledge. (1, 2)

An EBP is becoming an important issue in nursing, but it is poorly integrated into daily practice and its implementation is quite complex. Consider a process that consists of the following steps: 1) Translation of the clinical problem in the answered questions; 2) tracking with high efficiency in search of the best scientific evidence; 3) critical assessment of the findings regarding methodological quality; 4) integration of scientific evidence with clinical experience and patient values, with the implementation of findings in practice and; 5) evaluation of the implementation process and results. (2)

In the national scenario, one of the main challenges for evidence-based care is its implementation, since the expression of knowledge in action is considered a difficult process to be completed due to its complexity. (3)

In Brazil, the PBE movement is still not widespread in nursing work and in the process of training nurses. Few Brazilian institutions use a flow designed to guide their work processes in EBP, a movement that is occasionally found in the routine of health professionals. Still, with some resilience it has been used in professional practice, even if gradually. (3, 4)

The implementation of PBE in a hospital environment is considered a challenge. It is known that the standardization of assistance based on the best available evidence improves the results of patients, which goes against the concept of value-based medicine that has been widely disseminated. (2, 5)

Although the available literature on the subject points to positive attitudes of professional nurses and doctors regarding EBP, there is a disconnect between what these professionals believe and recognize with the actual implementation of EBP at the bedside. (5)

The main facilitating attitudes shared by nurses and doctors regarding EBP are: dedication of time to learn and practice, support from leadership, promotion of practice and easily accessible sources of evidence. (5)

These organizational and personal factors have a direct implication in the perception and development of this process in health institutions across the country.

When we analyze, for example, the individual beliefs of nurses working in the United States, the literature indicates that less than half, 41% (n = 656 / 1,564) agreed or strongly agreed that they knew how to implement PBE

sufficiently to make changes in practice clinic, and 44% (n = 701 / 1,564) were confident in their ability to implement. (5)

In Brazil, with regard to the individual beliefs of nurses, we found data from those who work in primary care, they recognize the importance and the need to perform EBP, however, the results indicated in the available literature revealed that the search for evidence is mostly based on clinical experience., patient preference and the use of opinions from colleagues in the profession or other institutions as the largest source of information to mediate clinical practice, as opposed to consultation with scientific sources. (4)

However, still exploring the Brazilian scenario, we find it a significant impediment to difficulties with the English language, as it is known that most of the relevant scientific productions in the area of health are produced and published in this language. (4)

We are experiencing a movement at the national level by some hospitals in the search for excellence in nursing practice. One of those responsible for this movement is the Magnet® recognition program that has encouraged institutions to seek the performance of nursing through PBE.

This program is aimed at hospital organizations and proposes to distinguish hospitals designated for high quality patient care and excellence in nursing care. (6)

Nursing research programs in organizations recognized as Magnet® have been growing, this growth is attributed to the requirements to achieve and maintain the designation that contribute to the science of nursing through research to discover new knowledge and implement PBE, in addition to training nurses. (6)

In comparison to unrecognized hospitals, nurses from Magnet® organizations report fewer difficulties associated with EBP, have more nurse research mentors designed to guide nurses at the bedside, with the development of a greater number of studies carried out by the clinical nurse as the main researcher, aligning three fundamental categories: research infrastructure, organizational research culture and construction of a research program for nursing. (6, 7)

Most of the hospital organizations recognized as Magnet® are located in North America. In Brazil, some hospitals intend or are on the journey (the period before the report is sent for the program to be evaluated) to achieve Magnet recognition in their institutions. To meet the recognition objectives, efforts are concentrated that directly involve increasing the levels of PBE implementation in these hospitals. (8)

In 2010 the institution where we operate was the first to join the Jornada Magnet and since 2012, several measures for the training of clinical nurses for greater scientific engagement have been implemented, an example was the hiring of a nurse researcher who works at the Research Institute, which has helped in the process of guiding and monitoring the scientific production of nurses and the institution's multidisciplinary team.

The initial diagnosis of the academic and scientific profile of clinical nurses at the institution revealed high heterogeneity of profiles, as well as some idiosyncrasies and beliefs in this population, which should be considered when implementing programs aimed at developing nursing research practices, as well as their Implementation. (9)

Basic level training programs with scientific methodology courses (8 hours), bibliographic research (regular library programs) and scientific writing (16 hours) have been developed over the years. For intermediate and advanced experience levels, courses in critical analysis of articles and scientific writing (40 hours) were also conducted.

In 2014, the Professional Master's Program in Institutional Nursing was created, which has played a fundamental role in the scientific training of clinical nurses. However, translating the knowledge generated into organizational clinical practice remains a challenge and this has been the responsibility of the Evidence-Based Practice Council, composed of nursing care leaders and the coordinators of the Magnet New Knowledge, Innovation and Improvements component, a nurse clinic and a researcher and professor, respectively, author and advisor of the present study.

This Council is designed to provide specialized guidance for clinical nurses, at all levels of training who want to gain experience in evidence-based practice, who work directly or indirectly in the care area, in conducting initiatives to elaborate and / or review protocols related to PBE directed to health care with quality and safety in several clinical outcomes.

Together with the PBE Council, clinical nurses have the guidance of the Library Service, which assists in the entire process of bibliographic search in databases. Even so, we have observed the degree of difficulties for this task and, mainly, for the critical analysis of scientific articles by clinical nurses.

The scenario of the Brazilian literature available on the topic of EBP presents mostly theoretical and reflective content, with few studies describing

changes in practice or interventions that support the dissemination of this practice in a hospital setting. (10)

Education strategies for the development of EBP focused on nursing leaders can be effective in decreasing the perception of the main difficulties for implementation, but it proved to be ineffective in expanding the skills of these leaders, leading to the reflection that focus on the formation of graduation of these professionals on this subject are important and relevant. (11)

The fact that we present the implementation of PBE as globally challenging, makes it necessary to investigate how the training of nurses has been developed by training institutions in this practice, in addition to discussions about the methodologies that best support this critical-reflective construction, the development of prospective studies that evaluate the impact of these methodologies in the training of professionals and the results in the quality of the assistance provided are essential to understand the best strategy to be adopted. (10, 11)

Taking into account the educational and training scenario as mentioned earlier, there are also gaps in the training of professionals.

The investigation of the knowledge, attitudes and practices of nursing students in implementing PBE, has shown that undergraduate nursing students do not have a high average knowledge score, and it is essential that colleges not only focus on education, but also assist students nurses to implement it in the patient care process. (12)

PBE education programs aimed at undergraduate nursing students are effective in improving knowledge, skills, attitudes and competencies, and are recommended to promote the necessary proficiency in PBE as part of professional training. On the other hand, how can we think of strategies aimed at clinical nurses who are already in the job market? (12, 13)

There is a gap in the production of studies on knowledge, attitudes and practices, and the difficulties in implementing PBE both in Brazil and in Latin America. This makes us reflect on what really happens and what is the collaboration for this scenario. (14)

The absence of a national model and facilitating instruments to assist this practice, considering that EBP is still under construction and growth in our environment, creates an even greater challenge for clinical nurses in our country, and that such reasoning may extend developing countries. (14)

In light of the above, this study aims to verify if the guide tools of the PBE model of the Johns Hopkins Nursing Evidence-based Practice, have a potential facilitator in the structuring and description of a PBE project conducted by Brazilian clinical nurses.

## 2. THEORETICAL FRAMEWORK

## 2.1 The Johns Hopkins model of evidence-based practice

The Johns Hopkins Evidence-Based Practice model resulted from the collaboration of nursing leaders in teaching and clinical practice at Johns Hopkins Hospital and Johns Hopkins University School of Nursing. The main objective of this model is to translate the best evidence for nurses who work at the bedside to use in care decisions. (15)

Your process has three steps called PET: Practical Questions, Evidence and Translation. This model is considered comprehensive, covering all important components of the PBE process. It is classified as individual, based on scientific and non-scientific evidence. (15)

In summary, the model includes tools divided into ten forms (Appendix 1) that serve as a guide to assist in the identification of an issue of care practice, to formulate the research question using terms appropriate to the search for evidence; seek, critically evaluate, summarize and classify the levels of evidence; and it also promotes the possibility of using non-scientific evidence (financial data, professional experience and patient preferences) for decision making. Based on that, the feasibility of applying the evidence is then determined, followed by the elaboration of an action plan for its translation, implementation of the change, evaluation and communication of results. (15, 16, 17)

The forms comprise:

 Appendix A\_PET Management Guide: Management guide with step by step description of the phases: practical question, evidence and translation, as well as spaces for projecting start dates, end of the project and those responsible for each step.

- Appendix B\_Question Development Tool: Brings key questions to help describe the problem raised for the construction of the initial PBE question, in addition to helping the beginning of the base for the search for evidence with the description of search terms and plan for measuring results. At the end of this form are the instructions that guide the completion.
- Appendix C\_Stakeholder Analysis: It has elements to characterize the stakeholders in the PBE project and their role in guaranteeing resources for implementing the action plan at the end of the project through the responsibilities of approvals, consultations and information.
- Appendix D\_Evidence Level and Quality Guide: Composed of guidelines and examples to help classify the levels of evidence that were found and their quality.
- Appendix E\_Research Appraisal Tool: This is a form made available to assist the user in the critical evaluation process of each evidence found. In this form we find elements to classify from the type of evidence, as to its quality according to the different types of study designs, such as, for example, quantitative, qualitative studies, systematic reviews, etc.
- Appendix F\_Non\_research Evidecen Appraisal Tool: The composition
  of this form assists in the classification of evidence considered "non-research",
  involves guidelines for clinical practices, consensus, expert opinions, in addition
  to the organizational experience of an institution.
- Appendix G\_Individual Evidence Tool: The purpose of this form is to document the key points of each evidence found in summary form, including

findings that help answer the clinical question and critical assessment data with level and quality classification, in order to prepare for the synthesis phase of this evidence.

- Appendix H Evidence Synthesis and Recommendation Tool: Proposes assistance in the description of a synthesis of the evidence findings, compiling the results that answer the PBE clinical question, brings the general classification and the final recommendation according to the level and quality of the evidence found, this recommendation may be strong, with convincing evidence and consistent results with solid indication for change of practice, or even little or no evidence with change of practice not indicated.
- Appendix I Action Planning Tool: This form has the purpose of guiding the construction of an action plan for planning the change in practice and guaranteeing a successful translation for all interested areas.
- Appendix J Dissemination Tool: Used at the end of the PBE project, it is a guide to the dissemination plan. It has fields for identifying the most appropriate communication methods for the defined target audience, whether individual, organizational or networks that may be interested in the results of the project, or that are part of the process of implementing the new practice.

In Brazil, the development of its own specific models is considered one of the main challenges, or the development of initiatives that portray the implementation and / or adaptation of the existing models proposed. (16)

## 2.2 The Magnet Model: New Knowledge, Innovations and Improvements Component

In the 1980s, studies by the American Academy of Nursing aimed to identify which were the main organizational characteristics that attract nurses, whose profile was considered to be a professional of excellence. (18)

The first research involving Magnet Hospitals was carried out in the 1980s, whose objective was to assess what characteristics these hospitals had that hindered or facilitated professional nursing practice. (18)

The results showed that some institutions had better results in recruiting and retaining the best nursing professionals. This study became a reference in the selection of the main attributes that underlie the direction patterns to determine the Magnet status. (18, 19)

The term "Magnet", which means "attraction" in the Portuguese language, has been used over the years to point out which hospitals are recognized by nurses as the best hospitals to work for. (18, 19)

In 1993, the Magnet Recognition Program® was established through the American Nurses Credentialing Center (ANCC), a subsidiary entity of the American Nursing Association (ANA) that is responsible for evaluating and recognizing health organizations that have Excellence Nursing Services. (20)

This program recommends actions that lead to the recognition and sharing of successful nursing practices and strategies.

Currently, only 10% of the 5,000 American hospitals are recognized, in addition to another 10 institutions located in Belgium, Jordan, Saudi Arabia, Lebanon, Australia, Canada and China. (8, 19, 21)

This recognition process is based on quality indicators and standards of good nursing practices from the American Nurses Association- ANA, the main areas evaluated are: (8, 19)

- 1) Transformational leadership The hospital environment has undergone reforms, including leadership, which were previously described as focused on stabilization and growth. Today's leaders are encouraged to transform the values, beliefs and behaviors of their institutions. (8)
- 2) Structure of empowerment Structures and processes developed by an influential leadership provide a transformative environment. It is observed that strong exemplary professional practice grows and that the results that are believed to be important are achieved through the living search for the institution's mission, vision and values. (8)
- 3) Exemplary professional practice the main essence of a Magnet institution is an exemplary professional practice in nursing. The objective of this component is more than the establishment of a strong professional practice, it is added what this professional practice can achieve. (8)
- 4) Empirical results Magnet institutions demonstrate results that must be categorized in terms of clinical results related to nursing practice: results of the workforce, results of patients, consumers and organizational results must be comparable with other institutions (subject to benchmarking). (8)
- 5) New knowledge, Innovation & Improvements Transformational leadership, trained professionals and exemplary practice are essential for institutions recognized as Magnet, but they are not the ultimate goals. These

institutions have an ethical and professional responsibility to contribute to patient care and the profession in terms of new knowledge, innovations and improvements. This component includes the design of new care models, the application of existing evidence, the search for new evidence and visible contributions to nursing science. This is the component to which the present study is related. (8)

The implementation of new knowledge, innovation and improvements brings reflections on how the clinical nurse who works in care and who is involved in research and EBP is able to implement changes in procedures and policies, positively impacting the outcomes resulting from nursing care to patients. (22)

It is framed and works side by side with another component previously described, called exemplary professional practice, which is able to demonstrate to the health community that the institution has achieved excellence and exemplary practice from the dedication of resources in order to continue on this path, acquiring new knowledge, using that knowledge to create innovations and improvements that help the patient, the institution where he works and the nursing profession. (22)

A Magnet® institution must support research and EBP, in addition to educating its nursing professionals in these elements. This is represented by the maintenance of researchers, educators and mentors who will assist in this process of supplying evidence and continuing education. (22, 23)

As part of the guidelines, institutions on their way to the Magnet® journey, they should initially consider some research practices such as:

differentiating research, PBE and improvement processes; incorporate that nurses who have researched and published their research evaluate and use the best results in their clinical practice; increase guidance on research and PBE projects; disseminate all the knowledge generated to internal and external forums. (22, 23)

## 2.3 The educational process in PBE: the four pillars of education

The approach to the mentoring process in the institution, both focused on research and on PBE, is based on the four pillars of education proposed by Jacques Delors: learn to know, learn to do, learn to live and learn to be, presented below. (24)

Learning to know, by combining a general culture, sufficiently broad, with the possibility of studying, in depth, a small number of subjects, that is: learning to learn, to benefit from the opportunities offered by lifelong education. (24)

Learning to do, in order to acquire not only a professional qualification, but, in a more comprehensive way, the competence that makes the person able to face numerous situations and to work as a team. In addition, learning to do in the context of different social or work experiences, whether spontaneously following the local or national context, or formally, thanks to the development of education alternated with work. (24)

Learning to live together, developing an understanding of the other and the perception of interdependencies - carrying out common projects and preparing to manage conflicts - while respecting the values of pluralism, mutual understanding and peace. (24)

Learning to be, in order to develop, as best as possible, the personality and to be in a position to act with an increasing capacity for self-autonomy, discernment and personal responsibility. For this purpose, education must take into account all the potential of each individual: memory, reasoning, aesthetic sense, physical capacities, ability to communicate. (24)

Thus, when applying the four pillars of education in our proposal for a facilitating model for PBE, we understand the four pillars as follows:

Learning to know: the search for evidence to establish the best nursing practices involves the development of skills in the search for information available in scientific publications, as well as the use of professional experience.

Learning to do evidence-based practice, in a broad sense, presupposes the use of a creative methodology of interaction with science that concretely proposes challenges to be overcome by seeking the best available evidence. Therefore, it presupposes knowing, analyzing and reflecting on the processes inherent to the elaboration of a PBE project. Knowing yourself in relation to the other influences how to do it, which is also essential for this process.

Learning to live is made possible, mainly, by the professional interaction that each nurse already develops in the health area, which enriches the teaching-learning process. However, when launching into the universe of EBP, nurses will go through one of the final phases that includes the dissemination of the findings of their search and application of the new practice based on the best evidence, this requires a broader capacity to live with other stakeholders involved in the studied process.

And, finally, learning to be comes through experience during and after the conclusion of a PBE project, characterized by the dissemination of the results found with all identified stakeholders. This stage is conducive to a reflective awakening for the nurse who developed the study regarding his relations with other nurses and managers during the activities developed, and planning future activities related to the development of new projects and professional development, thus awakening critical thinking to develop new clinical questions to search for evidence.

## 3. OBJECTIVES

## 3.1 General objective

Provide clinical nurses with tools to be used as a guide with a structured process in stages as a facilitator for the implementation of EBP projects in search of best practice in nursing processes.

## 3.2 Specific objectives

- 1) Check the adequacy of the authorized translation of the Portuguese language version of the Johns Hopkins Center for Evidence-Based Practice guide tools;
- 2) Analyze, from the perspective of the clinical nurse, if these tools are facilitators in the structuring and description of an EBP project;
- 3) Analyze, from the researcher's perspective, whether the PBE project met the requirements of: elaboration of a clinical question, bibliographic survey, critical evaluation of the evidence, summary of the evidence and elaboration of the dissemination plan;
- 4) Check if previous attitudes and knowledge regarding the implementation of PBE influence the structuring of a PBE project.

## 4. METHODOLOGY

## 4.1 Study type and location

Randomized study of educational intervention, comparative and prospective. The study will be carried out in the city of São Paulo at an Extra Large General Hospital that offers care from low to high complexity in several areas that include: critically ill patients unit, surgical medical clinic, oncology, surgical center, doctor's offices, various ambulatories and areas assistance support.

## 4.2 Population and sample

The target population of the study will be clinical nurses working in direct patient care, who meet the following inclusion and exclusion criteria.

## Inclusion criteria:

- Clinical nurse working at the bedside with at least two years of training in undergraduate nursing
- Intermediate self-reported English for reading

## Exclusion criteria:

 Having previously participated in a PBE project, the PBE council or research project, or even having a master's or doctor's degree.

For the recruitment of workshop participants, vacancies will be advertised through an invitation email addressed to the leaders of the institution, research location, with the proposed dates and times of PBE training, as well as the inclusion and exclusion criteria for selection. of the participants.

To calculate the sample, it will be taken into account that the variables of main interest in the study come from a questionnaire built by the researchers, so that we have no prior information about the distribution of the categories or the differences that we will find. With this data, 10 individuals in each group will be included in the study. After making comparisons between groups, if no evidence of differences is found, the observed data will be used to calculate the minimum sample size needed for a future study.

## 4.3 Study variables

Sociodemographic variables will be considered: age, training time and sex. Variable of interest: ease in structuring and describing an EBP project, from the perspective of the participating nurse and meeting the key elements of an EBP project, from the researcher's perspective.

Control variable: clinical nurse's practices, attitudes and prior knowledge about EBP.

## 4.4 Translation of tools

The translation of the Johns Hopkins Nursing Evidence-based Practice guide tools was authorized on 03/16/2018 by a representative of the Institute for Johns Hopkins Nursing documented through institutional email (Appendix 1).

The free translation was submitted for review by the Translation and Revision Service of the Einstein Integrated Library System, of the Albert Einstein Teaching and Research Institute, in February 2019.

The tools constitute a guiding guide and although this study is not about psychometric validation (as the tools do not measure any attribute), we chose to

present the authorized translation, to verify the adequacy of the translation by nurses who make up the Council of Practice Based on Evidence from Hospital Israelita Albert Einstein. For this purpose, a questionnaire will be used, prepared by the authors of this study, with closed questions: Questionnaire to check the adequacy of the authorized translation of the Portuguese language version of the Johns Hopkins PBE guide tools (Appendix 2).

The guide tools in the authorized version in Portuguese are: Appendix A - PET Management Guide, Appendix B - Question Development, Appendix C - Stakeholder Analysis, Appendix D - Evidence and Quality Level Guide, Appendix E - Assessment Tool Research Evidence Assessment, Appendix F - Non-Research Evidence Assessment Tool, Appendix G - Individual Evidence Tool, Appendix H - Evidence and Recommendations Synthesis Tool, Appendix I - Action Planning Tool, Appendix J - Dissemination tool. (Appendix 3).

For the verification phase of the adequacy of the authorized translation of the Portuguese language version of the guide tools, five specialists who work on the PBE Council will be invited. An email will be sent with the original versions in English and the translated versions of each tool into Brazilian Portuguese, as well as the questionnaire with closed questions and suggestions for improvements.

## 4.5 Educational strategies

Group A): will receive theoretical and practical training in PBE through a structured model workshop with themes related to the introduction to PBE, formulation of a practical question, bibliographic survey to search for evidence, critical analysis of evidence, classification of level and quality of information.

evidence, summarization and dissemination plan, with the final proposal of a practical class that aims to structure and describe an individual case through an exercise designed to go through the phases of a PBE project, as the basis for this exercise we will use a finalized and consolidated project, this will be used as a template for the exercise, the description of this exercise can be found in the programmatic content (Appendix 6). Group B): will receive the same training as group A, plus the presentation and availability of the Johns Hopkins Nursing Evidence-based Practice guide tools to be used in the practical class for the structuring and individual description of the PBE exercise case. The same theme of the case will be used in both groups.

Participants will be randomized and allocated to each of the educational intervention groups. For randomization, free software randomizer.org will be used.

## 4.6 Data collection

#### 4.6.1 Data collection instruments

The questionnaires that will be used in data collection are presented below.

- Questionnaire to check the adequacy of the authorized translation of the Portuguese language version of the Johns Hopkins PBE guide tools: Prepared by the researchers with a closed question about the intelligibility of the translation for the specialists, in addition to an open field for suggestions for changes. In case of inadequacy (which we define as less than four yes answers for the tools), we will make the changes mentioned by

the experts and submit the changed tools to a new evaluation by the experts. (Appendix 2).

- Evidence-Based Practice and Clinical Effectiveness Questionnaire (EBPQ): Validated and culturally adapted to the Brazilian Portuguese language in 2014 (25), it is a self-applicable instrument, considered important for assessing the use, opinions and knowledge of nurses about this practice. The instrument assesses attitudes, knowledge and implementation of PBE, uses a Likert-type scale with a score from one to seven in three domains: practice, attitudes and knowledge related to PBE. The objective of the applicability in this study will be for the variable of control of previous knowledge and through the analysis of the answers we will verify if the attitudes and previous knowledge in relation to the implementation of PBE influence in the structuring of a PBE project. (Annex 2).
- Questionnaire for the evaluation of the structuring process and description of an evidence-based practice project, from the perspective of the clinical nurse: Elaborated by the researchers considering the key elements of an EBP project (15) to verify the educational strategy to which was submitted facilitated the clinical nurse the process of elaborating an EBP project. The instrument consists of seven closed questions and one open for further comments. The closed questions are related to the description of a clinical question, ease in searching for evidence, understanding of scientific articles, ease in summarizing and classifying the levels of evidence, ease in describing the application of evidence and elaborating an action plan for disseminating the evidence.

evidence, in addition to the ease of going through all the phases of a PBE project in relation to the material offered during the workshop (with or without Johns Hopkins tools). (Appendix 4).

- Compliance verification questionnaire in structuring exercise and description of an evidence-based practice project from the researcher's perspective: Prepared by the researchers with five closed questions to verify compliance with the basic requirements and key elements of an EBP project. (Appendix 5). Definition criteria were established to standardize responses according to the researcher's observation. As a basis for determining this compliance in the questionnaire responses, we used as a reference the description of compliance parameters of the Joint Commission International published in the Joint Commission International survey process guide for clinical care program certification, 2014 (26), which comprises:

For yes and sufficient answers, compliance of or equal to 90%.

For partially sufficient and partially responses, compliance between 50 - 89%.

For no or insufficient responses, compliance is less than 49%.

For question 1: Was the participant able to elaborate a clinical question? One of the answers will be considered, yes or no. We will consider those who develop a clinical question according to the problem provided at the beginning of the exercise. It will be considered as an answer no, if the participant does not actually elaborate a clinical question, that is, an interrogative question about the problem received at the beginning of the exercise, or even, if the question elaborated is not using the problem provided as a basis.

For question 2: Regarding the survey of bibliographic articles, this was :.

One of the answers will be considered sufficient, partially sufficient or insufficient.

According to the compliance check, the values to be assigned and added to determine the response will be:

- a) Search terms previously consulted in the virtual health library in the section of health sciences descriptors for the search in the PubMed database 50% value
- b) Use of the two PubMed and CINAHL databases Value of 30% (Half the value will be considered if the search includes one of the two bases)
- c) Use of the advanced search module in the two databases Value of 20%. (Half the value will be considered if the advanced search is in one of the two bases)

**For question 3**: Regarding the classification of evidence according to the level of quality, was the participant able to carry out this classification? One of the answers will be considered: yes, partially or not.

According to the compliance check, the values to be assigned and added to determine the response will be:

a) Classification of the level of evidence I, II, III, IV and V by the participant in each of the articles provided for the exercise (total of 2 articles) - Value 20% for each article, total of 40%

- b) Evidence quality rating, A, B or C by the participant in each of the articles provided for the exercise (total of 2 articles) Value of 20% for each article, total of 40%
- c) Correct classification according to the exercise model Value of 10% for each article, total of 20%

**For question 4**: Was the participant able to elaborate a synthesis of the findings relating to the levels of evidence? One of the answers will be considered: yes, partially or not.

According to the compliance check, the values to be assigned and added to determine the response will be:

- Did the participant include the following points in the summary of the two articles provided for the exercise?
  - a) Type of study Value of 20%
  - b) Sample size Value of 20%
  - c) Summary of results and recommendations of the article Value of 20%
  - d) Classification of level of evidence and quality Value of 20%

Half of the value described (10%) will be considered if the participant presents a synthesis of only one of the two articles provided for the exercise in each of the topics from a) to d).

**For question 5**: Was the participant able to develop a dissemination plan for implementing the PBE project? One of the answers will be considered, yes, partially or not.

According to the compliance check, the values to be assigned and added to determine the response will be:

- Did the participant include the following points in the dissemination plan for implementing the PBE project?
- Project stakeholders Value of 20%
- Institution Leadership Value of 20%
- Department Leadership Value of 20%
- Front Line Team Value of 20%
- Dissemination methodology, example: online publication, presentation, meetings, etc. Value of 20%

The questionnaires will be inserted in the REDcap® digital platform, the participants will have access to the electronic resources notebook or tablet to insert their answers.

## 4.6.2 Operationalization of data collection

After recruiting the participants, workshops will be held, one for each group with a total workload of six hours divided into two consecutive days, lasting three hours each day. The first day will be theoretical and the second

day practical. The programmatic content of the workshops is described in the lesson plan. (Appendix 6).

The workshops with theoretical content and practical classes will be held in rooms of the Albert Einstein Hospital, preferably and according to availability at the Abram Szajman Health Education Center located at the Hospital Israelita Albert Einstein - Morumbi Unit.

All participants in both educational strategies will answer the same questionnaires.

Before the start of educational activities:

- Evidence-Based Practice and Clinical Effectiveness Questionnaire (EBPQ) (Annex 2).

At the end of the practical activity (second class):

- Evaluation Questionnaire on the structuring and description of an EBP project from the perspective of the clinical nurse (Appendix 4).

Subsequently, the case exercise performed by each participant during the practical class will be assessed by the researcher as to the conformity in the elaboration of the key phases of a PBE project through the questionnaire:

- Compliance verification questionnaire in the exercise of preparing a PBE project from the researcher's perspective (Appendix 5).

## 5. STATISTICAL ANALYSIS

The data collected will be described for EBP specialists and nurses in each group by means of absolute and relative frequencies for qualitative variables and by means and standard deviations or medians and quartiles for quantitative variables, depending on the observed sample distribution, which will be described by boxplot charts by groups. (21)

We will calculate the observed proportions of intelligibility for each translated tool and, in case of inadequacy (which we define as less than four yes answers for the tools), we will make the changes mentioned by the experts and submit the changed tools to a new evaluation by the experts.

For comparisons between groups of nurses considering qualitative variables, such as the items in the "questionnaire to assess the structuring and description of an evidence-based practice project from the perspective of the clinical nurse" and the "questionnaire to verify compliance in exercise of structuring and describing an evidence-based practice project from the researcher's perspective ", we will use chi-square tests or Fisher's exact tests and for comparisons considering quantitative variables we will use Student's t tests or Mann-Whitney tests, depending on sample distribution observed for the variables. (21)

The analyzes will be performed with the aid of the R package and considering a 5% significance level. (22)

## 6. ETHICAL ASPECTS

The project will be submitted to the Research Project Management System (SGPP) and the Research Ethics Committee (CEP) of the institution, the numbers of the approval protocols will be included in this work item.

In order to comply with the legal recommendations in force, the respective Terms of Free and Informed Consent (ICF) will be applied.

- Informed Consent Form (ICF) - SPECIALIST IN EVIDENCE-BASED PRACTICE

- Informed Consent Form (ICF) - NURSE.

Authorization was requested from the hospital's assistance director to conduct the study through the Term of Consent of the Area Managers, which met all institutional rules through the Term and Commitment of the Responsible Researcher in addition to the Term of Project Participants' Consent.

## **6. EXECUTION SCHEDULE**

| Schedule of Deliveries / Activities | | 2019 | | | 2020 | | | | | 2021 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Nov | Jan | Fev | Mar | Abr | Mai | Jun | 2°<br>Sem | Fev |
| 1 | SGPP Project Submission | Χ | | | | | | | | |
| 2 | Preparation of the content of the Workshops | | Х | | | | | | | |
| 3 | Submission of Johns Hopkins guides to expert judges | | | Х | | | | | | |
| 4 | Inclusion of participants | | | | Χ | Χ | | | | |
| 5 | PBE workshops | | | | | | Χ | Χ | | |
| 6 | Results analysis | | | | | | | | X | |
| 7 | Preparation of the final report | | | | | | | | Χ | Χ |

## 7. BIBLIOGRAPHIC REFERENCES

- 1. Pereira F, Salvi M, Verloo H. Beliefs, Knowledge, Implementation, and Integration of Evidence-Based Practice Among Primary Health Care Providers: Protocol for a Scoping Review. JMIR research protocols. 2017;6(8):e148.
- 2. Friesen-Storms JH, Moser A, van der Loo S, Beurskens AJ, Bours GJ. Systematic implementation of evidence-based practice in a clinical nursing setting: a participatory action research project. Journal of clinical nursing. 2015;24(1-2):57-68.
- 3. Danski MTR OG, Pedrolo E, Lind J, Johann D. A Importância da Prática Baseada em Evidências nos Processos de Trabalho do Enfermeiro. Cienc Cuid Saude 2017 Abr-Jun; 16(2). 2017.
- 4. Schneider LR, Pereira RPG, Ferraz L. A prática baseada em evidência no contexto da Atenção Primária à Saúde. Saúde debate. 2018;42(118):594-605.
- 5. Warren JI, McLaughlin M, Bardsley J, Eich J, Esche CA, Kropkowski L, et al. The Strengths and Challenges of Implementing EBP in Healthcare Systems. Worldviews on evidence-based nursing. 2016;13(1):15-24.
- 6. Pintz C, Zhou QP, McLaughlin MK, Kelly KP, Guzzetta CE. National Study of Nursing Research Characteristics at Magnet(R)-Designated Hospitals. The Journal of nursing administration. 2018;48(5):247-58.
- 7. Wilson M, Sleutel M, Newcomb P, Behan D, Walsh J, Wells JN, et al. Empowering nurses with evidence-based practice environments: surveying Magnet(R), Pathway to Excellence(R), and non-magnet facilities in one healthcare system. Worldviews on evidence-based nursing. 2015;12(1):12-21.
- 8. Magnet Recognition Program [homepage na internet]. ANCC Magnet Recognition Program® [acesso em 15/09/2019]. https://www.nursingworld.org/organizational-programs/magnet/.
- 9. Leão ER, Farah OG, Reis EAA, Barros CGd, Mizoi CS. Perfil acadêmico, crenças e autoeficácia em pesquisa de enfermeiros clínicos: implicações para o Programa de Pesquisa de Enfermagem de um Hospital na Jornada Magnet®. Einstein (São Paulo). 2013;11(4):507-13.

- 10. Camargo FC IH, Pereira GA, Souza RM, Garcia LAA, Monteiro DAT et al. . Estratégias para o ensino da prática baseada em evidências na formação de enfermeiros: Revisão Intergrativa. REFACS (online) 2018; 6(Supl 1):363-374.
- 11. Camargo FC PG, Iwamoto HH, Lorena LT, Goulart MB, Contim B. Oficinas para o desenvolvimento da prática baseada em evidências entre lideranças de enfermagem: estudo piloto. Rev Eletr Enf [Internet]. 2017;19:a50.
- 12. Ashktorab T, Pashaeypoor S, Rassouli M, Alavi-Majd H. Nursing Students' Competencies in Evidence-Based Practice and Its Related Factors. Nursing and midwifery studies. 2015;4(4):e23047.
- 13. Kim JS, Gu MO, Chang H. Effects of an evidence-based practice education program using multifaceted interventions: a quasi-experimental study with undergraduate nursing students. BMC medical education. 2019;19(1):71.
- 14. Camargo FC, Iwamoto HH, Galvão CM, Pereira GdA, Andrade RB, Masso GC. Competences and Barriers for the Evidence-Based Practice in Nursing: an integrative review. Rev Bras Enferm. 2018;71(4):2030-8.
- 15. Schaffer MA, Sandau KE, Diedrick L. Evidence-based practice models for organizational change: overview and practical applications. Journal of advanced nursing. 2013;69(5):1197-209.
- 16. Camargo FC, Iwamoto HH, Galvão CM, Monteiro DAT, Goulart MB, Garcia LAA. Modelos para a implementação da prática baseada em evidências na enfermagem hospitalar. Texto contexto enferm. 2018;26(4).
- 17. Center for Evidence-Based Practice [homepage na internet]. Johns Hopkins Medicine [acesso em 07/11/2019]. Disponível em: https://www.hopkinsmedicine.org/evidence-based-practice/ijhn\_2017\_ebp.html
- 18. Triolo PK, Scherer EM, Floyd JM. Evaluation of the Magnet Recognition Program. The Journal of nursing administration. 2006;36(1):42-8.
- 19. BARROS CGL, E. R.; REIS, E. A. A.; FARAH, O. G. . Excelência Assistencial: a Designação Magnet. Prática Hospitalar. 2012:São Paulo, p. 59 63.

- 20. McClure ML. Magnet hospitals: insights and issues. Nursing administration quarterly. 2005;29(3):198-201.
- 21. Aiken LH, Poghosyan L. Evaluation of "magnet journey to nursing excellence program" in Russia and Armenia. Journal of nursing scholarship: an official publication of Sigma Theta Tau International Honor Society of Nursing. 2009;41(2):166-74.
- 22. Barton SJ, Forster EK, Stuart ME, Patton AM, Rim JS, Torowicz DL. New knowledge, innovations, and improvement in a Magnet(R) Children's Hospital Cardiac Center. Journal of pediatric nursing. 2012;27(3):271-4.
- 23. Tinkham MR. The road to magnet: implementing new knowledge, innovations, and improvements. AORN journal. 2013;97(5):579-81.
- 24. Delors J. Learning: the treasure within; report to UNESCO of the International Commission on Education for the Twenty-first Century (highlights)2010.
- 25. Rospendowiski K, Alexandre NMC, Cornélio ME. Cultural adaptation to Brazil and psychometric performance of the "Evidence-Based Practice Questionnaire". Acta paul enferm. 2014;27(5):405-11.
- 26. Joint Commission International. Joint Commission International survey process guide for clinical care program certification. 3ª Edição, 2014

## 8. ATTACHMENTS:

## **ANNEX 1:**

PBE guiding tools for the Johns Hopkins Nursing Evidence-based Practice (original English versions).

2017 Appendix A PET Management Guide

2017\_Appendix B\_Question Development Tool

2017\_Appendix C\_Stakeholder Analysis

2017\_Appendix D\_Evidence Level and Quality Guide

2017\_Appendix E\_Research Appraisal Tool

2017\_Appendix F\_Non\_research Evidecen Appraisal Tool

2017 Appendix G Individual Evidence Tool

2017\_Appendix H Evidence Synthesis and Recommendation Tool

2017 Appendix I Action Planning Tool

2017 Appendix J Dissemination Tool

## 2017 Appendix A PET Management Guide



## **PRACTICE QUESTION**

- Step 1: Recruit interprofessional team
- Step 2: Define the problem
- Step 3: Develop and refine the EBP question
- Step 4: Identify stakeholders
- Step 5: Determine responsibility for project leadership
- Step 6: Schedule team meetings

## **EVIDENCE**

- Step 7: Conduct internal and external search for evidence
- Step 8: Appraise the level and quality of each piece of evidence
- Step 9: Summarize the individual evidence
- Step 10: Synthesize overall strength and quality of evidence
- Step 11: Develop recommendations for change based on evidence synthesis
  - Strong, compelling evidence, consistent results
  - Good evidence, consistent results
  - Good evidence, conflicting results
  - Insufficient or absent evidence

## **TRANSLATION**

Step 12: Determine fit, feasibility, and appropriateness of recommendation(s) for translation path

Step 13: Create action plan

Step 14: Secure support and resources to implement action plan

Step 15: Implement action plan

Step 16: Evaluate outcomes

Step 17: Report outcomes to stakeholders

Step 18: Identify next steps

Step 19: Disseminate findings

| Initial EDD Occasions | | | | | | | | | | | | |
|---|---|---|---|---|---|---|--|--|--|--|--|--|
| Initial EBP Question: | | | | | | | | | | | | |
| EBP Team Leader(s): EBP Team Members: | | | | | | | | | | | | |
| EDF Team Members. | Start | Days | End | Person | Milestone | Comment/ | | | | | | |
| Activities | Date | Required | Date | Assigned | | Resources<br>Required | | | | | | |
| PRACTICE QUESTION: | | | | | <del>-</del> | · | | | | | | |
| Step 1: Recruit interprofessional team | | | | | | | | | | | | |
| Step 2: Define the problem | | | | | | | | | | | | |
| Step 3: Develop and refine the EBP question | | | | | | | | | | | | |
| Step 4: Identify stakeholders | | | | | | | | | | | | |
| Step 5: Determine responsibility for project leadership | | | | | | | | | | | | |
| Step 6: Schedule team meetings | | | | | | | | | | | | |
| EVIDENCE: | | | | | | | | | | | | |
| Step 7: Conduct internal and external search for evidence | | | | | | | | | | | | |
| Step 8: Appraise the level and quality of each piece of evidence | | | | | | | | | | | | |
| Step 9: Summarize the individual evidence | | | | | | | | | | | | |
| Step 10: Synthesize overall strength and quality of evidence | | | | | | | | | | | | |
| Step 11: Develop recommendations for | | | | |
|---|---|---|--|--|
| change based on evidence | | | | |
| synthesis: | | | | |
| <ul> <li>Strong, compelling evidence,</li> </ul> | | | | |
| consistent results | | | | |
| <ul> <li>Good evidence, consistent</li> </ul> | | | | |
| results | | | | |
| <ul> <li>Good evidence, conflicting</li> </ul> | | | | |
| results | | | | |
| Insufficient or absent | | | | |
| evidence | | _ | | |
| TRANSLATION: | | | | |
| | ı ı | <del></del> | | |
| Step 12: Determine fit, feasibility, and | | | | |
| appropriateness of | | | | |
| recommendation(s) for | | | | |
| translation path | | | | |
| Step 13: Create action plan | | | | |
| 0: 11.0 | | | | |
| Step 14: Secure support and resources to | | | | |
| implement action plan | | | | |
| Step 15: Implement action plan | | | | |
| - Programme Prog | | | | |
| Step 16: Evaluate outcomes | | | | |
| Step 17: Report outcomes to stakeholders | | | | |
| Step 18: Identify next steps. | | | | |
| otop To: Identity Hext Steps. | | | | |
| Step 19: Disseminate findings. | | | | |

## 2017 Appendix B Question Development Tool

| 1. What is the problem? |
|---|
| 2. Why is the problem important and relevant? What would happen if it were not addressed? |
| 3. What is the current practice? |

| 4. How was the problem identified? (Check all that apply) | |
|---|---|
| □ Safety and risk-management concerns | □ Variations in practice within the setting |
| <ul> <li>Quality concerns (efficiency, effectiveness,<br/>timeliness, equity, patient-centeredness)</li> </ul> | <ul> <li>Variations in practice compared to community<br/>standard</li> </ul> |
| <ul> <li>Unsatisfactory patient, staff, or organizational</li> </ul> | □ Current practice that has not been validated |
| outcomes | □ Financial concerns |
| 5. What are the PICO components? | |
| P – (Patient, population, or problem) | |
| I – (Intervention) | |
| <b>C</b> – (Comparison with other interventions, if foreground qu | estion) |
| O – (Outcomes are qualitative or quantitative measures | s to determine the success of change) |
| 6. Initial EBP question ☐ Background ☐ Fo | reground |
| 7. List possible search terms, databases to sear | ch, and search strategies. |
| 8. What evidence must be gathered? (Check all | that apply) |
| □ Publications (e.g., EBSCOHost, PubMed, CINAHL, E | mbase) |
| ☐ Standards (regulatory, professional, community) | |
| □ Guidelines | |
| ☐ Organizational data (e.g., QI, financial data, local clin | ical expertise, patient/family preferences) |
| Position statements | |
| 9. Revised EBP question | |
| (Revisions in the EBP question may not be evident<br>be in the background question or a change from th | t until after the initial evidence review; the revision can e background to a foreground question) |
| 10. Outcome measurement plan | |

| What will we measure? (structure, process, outcome measure) | How will we measure it? (metrics are expressed as rate or percent) | How often will<br>we measure<br>it?<br>(frequency) | Where will we<br>obtain the<br>data? | Who will collect<br>the data? | o whom will we<br>report the<br>data? |
|---|---|---|---|---|---|

#### **Directions for Use of the Question Development Tool**

#### **Purpose**

This form is used to develop an answerable EBP question and to guide the team in the evidence search process. The question, search terms, search strategy, and sources of evidence can be revised as the EBP team refines the EBP question.

#### What is the problem, and why is it important?

Indicate why the project was undertaken. What led the team to seek evidence? Ensure that the problem statement defines the actual problem and does not include a solution. Whenever possible, quantify the extent of the problem. Validate the final problem description with practicing staff. It is important for the inter-professional team to take the time together to reflect, gather information, observe current practice, listen to clinicians, visualize how the process can be different or improved, and probe the problem description in order to develop a shared understanding of the problem.

#### What is the current practice?

Define the current practice as it relates to the problem. Think about current policies and procedures. Observe practices. What do you see?

#### How was the problem identified?

Check all the statements that apply.

#### What are the PICO components?

- **P** (patient, population, problem) e.g., age, sex, setting, ethnicity, condition, disease, type of patient, or population
- I (intervention) e.g., treatment, medication, education, diagnostic test, or best practice(s)
- **C** (comparison with other interventions or current practice for foreground questions; is not applicable for background questions, which identify best practice)
- **O** (outcomes) stated in measurable terms; may be a structure, a process, or an outcome measure based on the desired change (e.g., decrease in falls, decrease in length of stay, increase in patient satisfaction)

#### **Initial EBP question**

A starting question (usually a background question) that is often refined and adjusted as the team searches through the literature:

- Background questions are broad and are used when the team has little knowledge, experience, or expertise in the area of interest. Background questions are often used to identify best practices.
- Foreground questions are focused, with specific comparisons of two
  or more ideas or interventions. Foreground questions provide specific
  bodies of evidence related to the EBP question. Foreground questions
  often flow from an initial background question and literature review.

#### List possible search terms, databases to search, and search strategies.

Using PICO components and the initial EBP question, list search terms. Terms can be added or adjusted throughout the evidence search. Document the search terms, search strategy, and databases queried in sufficient detail for replication.

#### What evidence must be gathered?

Check the types of evidence the team will gather based on the PICO and initial EBP question.

#### **Revised EBP question**

Often, the question that you start with may not be the final EBP question. Back- ground questions can be refined or changed to a foreground question based on the evidence review. Foreground questions are focused questions that include specific comparisons and produce a narrower range of evidence.

#### Measurement plan

Measures can be added or changed as the review of the literature is completed and the translation planning begins:

- A measure is an amount or a degree of something, such as number of falls with injury. Each measure must be converted to a metric, which is calculated before and after implementing the change.
- Metrics let you know whether the change was successful. They have a numerator and a denominator and are typically expressed as rates or percent. For example, a metric for the measure falls-with-injury would be the number of falls with injury (numerator) divided by 1,000 patient days (denominator). Other examples of metrics include the number of direct care RNs (numerator) on a unit divided by the total number of direct care staff (denominator); the number of medication errors divided by 1,000 orders.

#### 2017 Appendix C Stakeholder Analysis

| 1. Identify the key stakeholders. | |
|---|---|
| <ul> <li>Manager or direct supervisor</li> <li>Finance department</li> <li>Vendors</li> <li>Patients and/or families; patient and family advisory committee</li> </ul> | <ul> <li>Organizational leaders</li> <li>Interdisciplinary colleagues (e.g. physicians, nutritionists, respiratory therapists, or OT/PT)</li> <li>Administrators</li> <li>Other units or departments</li> </ul> |
| □ Professional organizations | □ Others: |
| □ Committees | |
| 2. Stakeholder roles and responsibilities. | |
| (The stakeholder roles—which include Responsibility, Consult, Approval, and Inform and their corresponding | |
| responsibilities, described here—guide completion of the | • |

| Responsibilit | ty | Consult | |
|---|---|---|---|
| · · | etes identified tasks<br>mending authority | <ul><li>Provides input (e.g., subject matter experts)</li><li>No decision-making authority</li></ul> | |
| Approval | | Inform | |
| <ul><li>Signs off on recommendations</li><li>May veto</li></ul> | | <ul><li>Notified of progress and changes</li><li>No input on decisions</li></ul> | |
| Project tasks | Stakeholder name | Stakeholder name | Stakeholder name |
| ., | Stakeholder role | Stakeholder role | Stakeholder role |

#### Directions for Use of the Stakeholder Analysis Tool

#### **Purpose**

This form is used to identify key stakeholders. Key stakeholders are persons, groups, or departments in the organization that have an interest in, or concern about, your project and/or may assist you in securing resources to implement your action plan. Involve stakeholders early in the process to ensure their buy-in for implementation.

Because stakeholders may change at different steps of the process, we recommend that you review this form as you proceed from step to step in your action plan.

#### Definition

Stakeholders are "persons or groups that have a vested interest in a clinical [or nonclinical] decision and the evidence that supports that decision" (AHRQ, 2014).

#### Identify the key stakeholders

Identify the 5–7 key stakeholders who can most affect, or who will be most affected by, the project, actions, objectives, or change and who can influence the success of the translation work. Key stakeholders are individuals or groups who:

- Make decisions about the project
- Approve the project or aspects of the project
- Serve as subject matter experts
- Provide resources such as support, policy changes, resources, and time

#### Stakeholder analysis

It is helpful to consider which of the four roles each stakeholder may play in your action planning and translation work. The possible roles are:

- Responsibility
- Approval
- Consult
- Inform

Remember that one stakeholder may fill different roles, depending on the action. Completion of the Stakeholder Analysis Tool will help clarify roles and responsibilities. The descriptions of responsibilities for each role provided on the form will be helpful in this process.

References: Agency for Healthcare Research and Quality. (2014) .Stakeholder Guide 2014 .Retrieved from www.effectivehealthcare.ahrq.gov.AHRQ Publication No. 14-EHC010-EF. Replaces Publication No. 11-EHC069-EF

## 2017 Appendix D Evidence Level and Quality Guide

#### Appendix D

Evidence Level and Quality Guide

| Evidence Levels | Quality Ratings |
|---|---|
| Level I | QuaNtitative Studies |
| Experimental study, randomized controlled trial (RCT) | A <u>High quality</u> : Consistent, generalizable results; sufficient sample size for the study design; adequate control; definitive conclusions; consistent recommendations based on comprehensive literature review that includes thorough reference to scientific evidence. |
| Explanatory mixed method design that includes only a level I quaNtitative study | B <u>Good quality</u> : Reasonably consistent results; sufficient sample size for the study design; some control, fairly definitive conclusions; reasonably consistent recommendations based on fairly comprehensive literature review that includes some reference to scientific evidence. |
| Systematic review of RCTs, with or without meta-<br>analysis | C <u>Low quality or major flaws</u> : Little evidence with inconsistent results; insufficient sample size for the study design; conclusions cannot be drawn. |
| Level II | QuaLitative Studies |
| Quasi-experimental study | No commonly agreed-on principles exist for judging the quality of qualitative studies. It is a subjective |
| Explanatory mixed method design that includes | process based on the extent to which study data contributes to synthesis and how much information is known about the researchers' efforts to meet the appraisal criteria. |
| only a level II quaNtitative study | Formeta-synthesis, there is preliminary agreement that quality assessments of individual studies should be |
| Systematic review of a combination of RCTs and<br>quasi-experimental studies, or quasi- | made before synthesis to screen out poor-quality studies <sup>1</sup> , |
| experimental studies only, with or without meta- | A/B <u>High/Good quality</u> is used for single studies and meta-syntheses <sup>2</sup> . |
| analysis | The report discusses efforts to enhance or evaluate the quality of the data and the overall inquiry in<br>sufficient detail; and it describes the specific techniques used to enhance the quality of the inquiry.<br>Evidence of some or all of the following is found in the report: |
| Level III<br>Nonexperimental study | <ul> <li>Transparency: Describes how information was documented to justify decisions, how data were<br/>reviewed by others, and how themes and categories were formulated.</li> </ul> |
| Systematic review of a combination of RCTs, quasi-experimental and nonexperimental studies, | <ul> <li>Diligence: Reads and rereads data to check interpretations; seeks opportunity to find multiple<br/>sources to comoborate evidence.</li> </ul> |
| or nonexperimental studies only, with or without | <ul> <li>Verification: The process of checking, confirming, and ensuring methodologic coherence.</li> </ul> |
| meta-analysis | <ul> <li>Self-reflection and scrutiny: Being continuously aware of how a researcher's experiences,<br/>background, or prejudices might shape and bias analysis and interpretations.</li> </ul> |
| Exploratory, convergent, or multiphasic mixed<br>methods studies | <ul> <li>Participant-driven inquiry: Participants shape the scope and breadth of questions; analysis and</li> </ul> |
| Explanatory mixed method design that includes | interpretation give voice to those who participated. |
| only a level III quaNtitative study | <ul> <li>Insightful interpretation: Data and knowledge are linked in meaningful ways to relevant literature.</li> </ul> |
| QuaLitative study Meta-synthesis | C <u>Low quality</u> studies contribute little to the overall review of findings and have few, if any, of the features listed for high/good quality. |

#### Appendix D

**Evidence Level and Quality Guide** 

| Evidence Levels | Quality Ratings |
|---|---|
| Level IV Opinion of respected authorities and/or nationally recognized expert committees or consensus panels based on scientific evidence Includes: • Clinical practice guidelines • Consensus panels/position statements | A High quality: Material officially sponsored by a professional, public, or private organization or a government agency; documentation of a systematic literature search strategy; consistent results with sufficient numbers of well-designed studies; criteria-based evaluation of overall scientific strength and quality of included studies and definitive conclusions; national expertise clearly evident; developed or revised within the past five years B Good quality: Material officially sponsored by a professional, public, or private organization or a government agency; reasonably thorough and appropriate systematic literature search strategy; reasonably consistent results, sufficient numbers of well-designed studies; evaluation of strengths and limitations of included studies with fairly definitive conclusions; national expertise clearly evident; developed or revised within the past five years C Low quality or major flaws: Material not sponsored by an official organization or agency; undefined, poorly defined, or limited literature search strategy; no evaluation of strengths and limitations of included studies, insufficient evidence with inconsistent results, conclusions cannot be drawn; not revised within the past five years |
| Level V Based on experiential and nonresearch evidence Includes: Integrative reviews Literature reviews Quality improvement, program, or financial evaluation Case reports Opinion of nationally recognized expert(s) based on experiential evidence | Organizational Experience (quality improvement, program or financial evaluation) A High quality: Clear aims and objectives; consistent results across multiple settings; formal quality improvement, financial, or program evaluation methods used; definitive conclusions; consistent recommendations with thorough reference to scientific evidence B Good quality: Clear aims and objectives; consistent results in a single setting; formal quality improvement, financial, or program evaluation methods used; reasonably consistent recommendations with some reference to scientific evidence C Low quality or major flaws: Unclear or missing aims and objectives; inconsistent results; poorly defined quality improvement, financial, or program evaluation methods; recommendations cannot be made Integrative Review, Literature Review, Expert Opinion, Case Report, Community Standard, Clinician Experience, Consumer Preference A High quality: Expertise is clearly evident; draws definitive conclusions; provides scientific rationale; thought leader(s) in the field B Good quality: Expertise appears to be credible; draws fairly definitive conclusions; provides logical argument for opinions C Low quality or major flaws: Expertise is not discernable or is dubious; conclusions cannot be drawn |

1 https://www.york.ac.uh/cd/BysRev/ISSU/WebHc by/e\_4\_ASSESSMENT\_OF\_QUAUTATIVE\_MESEARCH Non-2 Adopted from Polk & Seek (2017).

# 2017 Appendix E Research Appraisal Tool

| Evidence level and quality rating: | |
|---|---|
| Article title: | Number: |
| Author(s): | Publication date: |
| Journal: | |
| Setting: | Sample (composition and size): |
| Does this evidence address my EBP question? | |
| ☐ Yes<br>☐ No- <i>Do not proceed with appraisal o</i> | of this evidence |
| In the second or | |
| Is this study: | |
| QuaNtitative (collection, analysis, and reporting of numerical data) Measurable data (how many; how much; or how often) used to formulate facts, uncover patterns in research, and generalize results from a larger sample population; provides observed effects of a program, problem, or condition, measured precisely, rather than through researcher interpretation of data. Common methods are surveys, face-to-face structured interviews, observations, and reviews of records or documents. Statistical tests are used in data analysis. | |
| Go to <b>Section I: QuaNtitative</b> | |
| Qualitative (collection, analysis, and reporting of narrative data) Rich narrative documents are used for uncovering themes; describes a problem or condition from the point of view of those experiencing it. Common methods are focus groups, individual interviews (unstructured or semi structured), and participation/observations. Sample sizes are small and are determined when data saturation is achieved. Data saturation is reached when the researcher identifies that no new themes emerge and redundancy is occurring. Synthesis is used in data analysis. Often a starting point for studies when little research exists; may use results to design empirical studies. The researcher describes, analyzes, and interprets reports, descriptions, and observations from participants. Go to Section II: Qualitative | |
| ☐ Mixed methods (results reported | both numerically and narratively) |
| Both quaNtitative and quaLitative methods are used combination, provides a better understanding of reseasing sample sizes vary based on methods used. Data of quaNtitative and quaLitative data in a single study or can influence stages in the research process. | in the study design. Using both approaches, in arch problems than using either approach alone. collection involves collecting and analyzing both |
| Go to Section I for QuaNtitative components a | nd Section II for QuaLitative components |

| Section I: QuaNtitative | | |
|---|---|---|
| Level of Evidence (Study Design) | | |
| A Is This a report of a single research study? | □ Yes | □No<br><b>Go to B</b> |
| 1. Was there manipulation of an independent variable? | □ Yes | □ No |
| 2. Was there a control group? | □ Yes | □ No |
| Were study participants randomly assigned to the intervention and control groups? | □ Yes | □ No |
| Yes to questions 1, 2, and 3, this is a randomized controlled trial (RCT) experimental study. | LEVEL I | |
| Yes to questions 1 and 2 and No to question 3 or Yes to question 1 and No to questions 2 and 3, this is quasi-experimental. (Some degree of investigator control, some manipulation of an independent variable, lacks random assignment to groups, and may have a control group). | | |
| No to questions 1, 2, and 3, this is nonexperimental. (No manipulation of independent variable; can be descriptive, comparate correlational; often uses secondary data). | LEVEL III | |
| Study Findings That Help Answer the EBP Question | | |
| Complete the Appraisal of QuaNtitative Research Studies section | | |

| Is this a summary of multiple sources of research evidence? | □ Yes<br>Continue | □ No<br>Use Appendix F |
|---|---|---|
| 1. Does it employ a comprehensive search strategy and rigorous appraisal method? If this study includes research, nonresearch, and experiential evidence, it is an integrative review (see Appendix F). | | □ No<br>Use Appendix F |
| <ol><li>For systematic reviews and systematic reviews with meta-<br/>(see descriptions below):</li></ol> | analysis | |
| a. Are all studies included RCTs? | | LEVEL I |
| b. Are the studies a combination of RCTs and q or quasi-experimental only? | uasi-experimental, | LEVEL II |
| c. Are the studies a combination of RCTs, quas nonexperimental, or non- experimental only? | | LEVEL III |
| A <u>systematic review</u> employs a search strategy and a rigorous appraisal method, but does not generate an effect size. A <u>meta-analysis</u> , or systematic review with meta-analysis, combines and analyzes results from studies to generate a new statistic: the effect size. | | |
| Study Findings That Help Answer the EBP Question Complete the Appraisal of Systematic Review (With or Without) | out a Meta-Analysis) s | ection |
| Complete the <b>Appraisal of Systematic Review</b> (With or Witho | iut a ivieta-Analysis) se | ecuon |

| Appraisal of QuaNtitative Research Studies | | | |
|---|---|---|---|
| Does the researcher identify what is known and not known about the problem and how the study will address any gaps in knowledge? | □ Yes | □ No | |
| Was the purpose of the study clearly presented? | □ Yes | □ No | |
| Was the literature review current (most sources within the past five years or a seminal study)? | □ Yes | □ No | |
| Was sample size sufficient based on study design and rationale? | □ Yes | □ No | |
| <ul> <li>If there is a control group:</li> <li>Were the characteristics and/or demographics similar in both the control and intervention groups?</li> </ul> | □ Yes | □ No | N/A |
| <ul> <li>If multiple settings were used, were the settings<br/>similar?</li> </ul> | □ Yes | □ No | N/A |
| <ul> <li>Were all groups equally treated except for the<br/>intervention group(s)?</li> </ul> | □ Yes | □ No | N/A |
| Are data collection methods described clearly? | □ Yes | □ No | |
| Were the instruments reliable (Cronbach's [alpha] > 0.70)? | □ Yes | □ No | N/A |
| Was instrument validity discussed? | □ Yes | □ No | N/A |
| If surveys or questionnaires were used, was the response rate > 25%? | □ Yes | □ No | N/A |
| Were the results presented clearly? | □ Yes | □ No | |
| If tables were presented, was the narrative consistent with the table content? | □ Yes | □ No | N/A |
| Were study limitations identified and addressed? | □ Yes | □ No | |
| Were conclusions based on results? | □ Yes | □ No | |
| Go to Quality Rating for QuaNtitative Studies section | | | |

| Appraisal of Systematic Review (With or Without Meta-Analysis) | | |
|---|---|---|
| Were the variables of interest clearly identified? | □ Yes | □ No |
| Was the search comprehensive and reproducible? • Key search terms stated | □ Yes | □ No |
| Multiple databases searched and identified | □ Yes | □ No |
| Inclusion and exclusion criteria stated | □ Yes | □ No |
| Was there a flow diagram that included the number of studies eliminated at each level of review? | □ Yes | □ No |
| Were details of included studies presented (design, sample, methods, results, outcomes, strengths, and limitations)? | □ Yes | □ No |
| Were methods for appraising the strength of evidence (level and quality) described? | □ Yes | □ No |
| Were conclusions based on results? | □ Yes | □ No |
| Results were interpreted | □ Yes | □ No |
| Conclusions flowed logically from the interpretation and systematic review question | □ Yes | □ No |
| Did the systematic review include a section addressing limitations <u>and</u> how they were addressed? | □ Yes | □ No |
| Complete Quality Rating for QuaNtitative Studies section | | |

#### **Quality Rating for QuaNtitative Studies**

Circle the appropriate quality rating below:

- A High quality: Consistent, generalizable results; sufficient sample size for the study design; adequate control; definitive conclusions; consistent recommendations based on comprehensive literature review that includes thorough reference to scientific evidence.
- **B Good quality**: Reasonably consistent results; sufficient sample size for the study design; some control, and fairly definitive conclusions; reasonably consistent recommendations based on fairly comprehensive literature review that includes some reference to scientific evidence.
- **C Low quality or major flaws**: Little evidence with inconsistent results; insufficient sample size for the study design; conclusions cannot be drawn.

| Section II: QuaLitative | | |
|---|---|---|
| Level of Evidence (Study Design) | | |
| A Is this a report of a single research study? | □ Yes<br>go to Level III | □ No<br>go to II B |
| Study Findings That Help Answer the EBP Question | | |
| Complete Appraisal of Single QuaLitative Research Study section | | |

| Appraisal of a Single QuaLitative Research Study | | |
|---|---|---|
| Was there a clearly identifiable and articulated: • Purpose? | □ Yes | □No |
| Research question? | □ Yes | □ No |
| Justification for method(s) used? | □ Yes | □ No |
| Phenomenon that is the focus of the research? | □ Yes | □No |
| Were study sample participants representative? | □ Yes | □ No |
| Did they have knowledge of or experience with the research area? | □ Yes | □ No |
| Were participant characteristics described? | □ Yes | □ No |
| Was sampling adequate, as evidenced by achieving saturation of data? | □ Yes | □ No |
| Data analysis: | | |
| <ul> <li>Was a verification process used in every step by checking and confirming<br/>with participants the trustworthiness of analysis and interpretation?</li> </ul> | □Yes | □No |
| <ul> <li>Was there a description of how data were analyzed (i.e., method), by<br/>computer or manually?</li> </ul> | □ Yes | □No |
| Do findings support the narrative data (quotes)? | □Yes | □ No |
| Do findings flow from research question to data collected to analysis undertaken? | □ Yes | □No |
| Are conclusions clearly explained? | □ Yes | □No |
| Go to Quality Rating for Qualitative Studies section | | |

| В | For summaries of multiple quaLitative research studies (meta-synthesis), was a comprehensive search strategy and rigorous appraisal method used? | □ Yes<br>Level III | □ No<br>go to <b>Appendix F</b> |
|---|---|---|---|
| Study | Findings That Help Answer the EBP Question | | |
| Coi | mplete the Appraisal of Meta-Synthesis Studies section | | |

| Appraisal of Meta-Synthesis Studies | | |
|---|---|---|
| Were the search strategy and criteria for selecting primary studies clearly defined? | □ Yes | □No |
| Were findings appropriate and convincing? | □ Yes | □ No |
| Was a description of methods used to: • Compare findings from each study? | □ Yes | □No |
| Interpret data? | □ Yes | □No |
| Did synthesis reflect: | □ Yes | □No |
| New insights? | □ Yes | □ No |
| Discovery of essential features of phenomena? | □ Yes | □No |
| A fuller understanding of the phenomena? | □ Yes | □ No |
| Was sufficient data presented to support the interpretations? | □ Yes | □ No |
| Complete the Quality Rating for Qualititative Studies section | | |

#### **Quality Rating for QuaLitative Studies**

Circle the appropriate quality rating below:

No commonly agreed-on principles exist for judging the quality of quaLitative studies. It is a subjective process based on the extent to which study data contributes to synthesis and how much information is known about the researchers' efforts to meet the appraisal criteria.

For meta-synthesis, there is preliminary agreement that quality assessments should be made before synthesis to screen out poor-quality studies<sup>1</sup>.

A/B <u>High/Good quality</u> is used for single studies and meta-syntheses<sup>2</sup>.

The report discusses efforts to enhance or evaluate the quality of the data and the overall inquiry in sufficient detail; and it describes the specific techniques used to enhance the quality of the inquiry.

Evidence of some or all of the following is found in the report:

- **Transparency**: Describes how information was documented to justify decisions, how data were reviewed by others, and how themes and categories were formulated.
- **Diligence**: Reads and rereads data to check interpretations; seeks opportunity to find multiple sources to corroborate evidence.
- **Verification**: The process of checking, confirming, and ensuring methodologic coherence.
- **Self-reflection and self-scrutiny**: Being continuously aware of how a researcher's experiences, background, or prejudices might shape and bias analysis and interpretations.
- Participant-driven inquiry: Participants shape the scope and breadth of questions; analysis and interpretation give voice to those who participated.
- Insightful interpretation: Data and knowledge are linked in meaningful ways to relevant literature.
- **C** <u>Lower-quality</u> studies contribute little to the overall review of findings and have few, if any, of the features listed for High/Good quality.

# Section III: Mixed Methods Level of Evidence (Study Design) You will need to appraise both the quaNtitative and quaLitative parts of the study independently, before appraising the study in its entirety. 1. Evaluate the quaLitative part of the study using Section I. Insert here the level of evidence and overall quality for this part: 2. Evaluate the quaLitative part of the study using Section II. Level Quality

| Insert here the level of evidence and overall quality for this part: | | | |
|---|---|---|---|
| 3. To determine the level of evidence, circle the appropriate study design: | | | |
| <ul> <li>Explanatory sequential designs collect quaNtitative data first, followed by the opurpose is to explain quaNtitative results using quaLitative findings. The level is level of the quaNtitative part.</li> </ul> | | | |
| <ul> <li>Exploratory sequential designs collect quaLitative data first, followed by the quenting purpose is to explain quaLitative findings using the quaNtitative results. The level the level of the quaLitative part, and it is always Level III.</li> </ul> | | | |
| <ul> <li>Convergent parallel designs collect the quaLitative and quaNtitative data conceptoriding a more complete understanding of a phenomenon by merging both data Level III.</li> </ul> | | | |
| <ul> <li>Multiphasic designs collect quaLitative and quaNtitative data over more than of informing the next phase. These designs are Level III.</li> </ul> | ne phase | e, with ea | ach phase |
| Study Findings That Help Answer the EBP Question | | | |
| Use the Appraisal of Mixed Methods Studies section | | | |
| Appraisal of Mixed Methods Studies <sup>3</sup> | | | |
| Was the mixed-methods research design relevant to address the quaNtitative and quaLitative research questions (or objectives)? | □ Yes | □ No | □ N/A |
| Was the research design relevant to address the quaNtitative and quaLitative aspects of the mixed-methods question (or objective)? | □ Yes | □ No | □ N/A |
| For convergent parallel designs, was the integration of quaNtitative and quaLitative data (or results) relevant to address the research question or objective? | □ Yes | □ No | □ N/A |

Go to Quality Rating for Mixed-Method Studies section

results) sufficiently addressed?

For convergent parallel designs, were the limitations associated with the integration (for example, the divergence of quaLitative and quaNtitative data or

□ No

□ Yes

□ N/A

| Appraisal of Meta-Synthesis Studies | | |
|---|---|---|
| Were the search strategy and criteria for selecting primary studies clearly defined? | □ Yes | □No |
| Were findings appropriate and convincing? | □Yes | □No |
| Was a description of methods used to: • Compare findings from each study? | □ Yes | □No |
| Interpret data? | □Yes | □No |
| Did synthesis reflect: | □Yes | □No |
| New insights? | □Yes | □No |
| Discovery of essential features of phenomena? | □ Yes | □No |
| A fuller understanding of the phenomena? | □Yes | □ No |
| Was sufficient data presented to support the interpretations? | □Yes | □No |
| Complete the Quality Rating for Qualtitative Studies section | | |

#### **Quality Rating for Mixed-Methods Studies**

Circle the appropriate quality rating below

- A <u>High quality</u>: Contains high-quality quaNtitative and quaLitative study components; highly relevant study design; relevant integration of data or results; and careful consideration of the limitations of the chosen approach.
- **B** <u>Good quality</u>: Contains good-quality quaNtitative and quaLitative study components; relevant study design; moderately relevant integration of data or results; and some discussion of limitations of integration.
- **C** <u>Low quality or major flaws</u>: Contains low quality quaNtitative and quaLitative study components; study design not relevant to research questions or objectives; poorly integrated data or results; and no consideration of limits of integration.

# 2017 Appendix F Non research Evidecen Appraisal Tool

| Evidence level and quality rating: | | | | | |
|---|---|---|---|---|---|
| Article title: | Number: | | | | |
| Author(s): | Publication dat | te: | | | |
| Journal: | | | | | |
| Setting: Sample (composition and size): | | | | | |
| Does this evidence address my EBP question? ☐ Yes ☐ No- Do not proceed with appraisal of this e | evidence | | | | |
| □ Clinical Practice Guidelines LEVEL IV Systematically developed recommendations from nationally evidence or expert consensus panel □ Consensus or Position Statement LEVEL IV Systematically developed recommendations, based on rescopinion, that guide members of a professional organization concern | earch and na | tiona | ally recog | nized | expert |
| Are the types of evidence included identified? | | | Yes | | No |
| Were appropriate stakeholders involved in the developmer recommendations? | nt of | | Yes | | No |
| • Are groups to which recommendations apply and do not ap<br>stated? | oply clearly | | Yes | | No |
| Have potential biases been eliminated? | | | Yes | | No |
| Does each recommendation have an identified level of evid | dence stated? | | Yes | | No |
| Are recommendations clear? | | | Yes | | No |
| Findings That Help Answer the EBP Question | | | | | |
| Complete the corresponding quality rating section. | | | | | |

| □ Literature review LEVEL V Summary of selected published literature including scientific and nonso organizational experience and opinions of experts | entif | ic such a | as re | ports of |
|---|---|---|---|---|
| □ Integrative review LEVEL V Summary of research evidence and theoretical literature; analyzes, comin the selected literature | ıpare | s themes | s, not | es gaps |
| Is subject matter to be reviewed clearly stated? | | Yes | | No |
| <ul> <li>Is literature relevant and up-to-date (most sources are within the past five<br/>years or classic)?</li> </ul> | | Yes | | No |
| Of the literature reviewed, is there a meaningful analysis of the conclusions across the articles included in the review? | | Yes | | No |
| Are gaps in the literature identified? | | Yes | | No |
| Are recommendations made for future practice or study? | | Yes | | No |
| Complete the corresponding quality rating section. | | | | |
| □ Expert opinion LEVEL V Opinion of one or more individuals based on clinical expertise | | | | |
| <ul> <li>Has the individual published or presented on the topic?</li> </ul> | | Yes | | No |
| Is the author's opinion based on scientific evidence? | | Yes | | No |
| Is the author's opinion clearly stated? | | Yes | | No |
| Are potential biases acknowledged? | | Yes | | No |
| Findings That Help Answer the EBP Question | | | | |
| Complete the corresponding quality rating section. | | | | |

| Org | janizational Experience | | | | | |
|---|---|---|---|---|---|---|
| | Quality improvement LEVEL V Cyclical method to examine workflows, processes, or system | ns with | a specific o | rganizat | tion | |
| | □ Financial evaluation LEVEL V Economic evaluation that applies analytic techniques to identify, measure, and compare the cost and outcomes of two or more alternative programs or interventions | | | | | cost and |
| | Program evaluation LEVEL V Systematic assessment of the processes and/or outcomes of quaNtitative and quaLitative methods | of a prog | gram; can in | volve b | oth | |
| Setting | g: | Sample | Size/Compo | osition: | | |
| • | Was the aim of the project clearly stated? | [ | ⊐Yes | □ N | lo | |
| • | Was the method fully described? | [ | ⊐Yes | □N | lo | |
| • | Were process or outcome measures identified? | [ | ⊐Yes | ΩN | lo | |
| • | Were results fully described? | [ | ⊐ Yes | □N | lo | |
| • | Was interpretation clear and appropriate? | [ | ⊐ Yes | | lo | |
| • | Are components of cost/benefit or cost effectiveness analysis described? | J | ⊐Yes | οN | lo | □ N/A |
| Findir | ngs That Help Answer the EBP Question | | | | | |
| Coi | mplete the corresponding quality rating section. | | | | | |
| _ | Case report LEVEL V In-depth look at a person or group or another social unit | | | | | |
| | ■ Is the purpose of the case report clearly stated? | | □ Ye: | s | | □ No |
| | ■ Is the case report clearly presented? | | □ Ye: | s | | □No |

• Are the findings of the case report supported by relevant theory or research?

□ No

□ Yes

| • Are the recommendations clearly stated and linked to<br>findings? | o the | □Yes | □ No |
|---|---|---|---|
| Findings That Help Answer the EBP Question | | | |
| Complete the corresponding quality rating. | | | |
| g quantity and g | | | |
| Community standard, clinician experience, or consu | mer prefe | rence LEVEL V | |
| Community standard: Current practice for comparab | le settings i | n the community | |
| □ Clinician experience: Knowledge gained through pra | actice expe | rience | |
| Consumer preference: Knowledge gained through life expe | rience | | |
| Information Source(s) | | Number of Sources | |
| Source of information has credible experience | □Yes | □No | □ N/A |
| Opinions are clearly stated | □Yes | □No | □ N/A |
| Evidence obtained is consistent | □Yes | □No | □ N/A |
| Findings That Help You Answer the EBP Question | | | |
| Complete the corresponding quality rating section. | | | |

#### Quality Rating for Clinical Practice Guidelines, Consensus, or Position Statements (Level IV)

#### A High quality

Material officially sponsored by a professional, public, or private organization or a government agency; documentation of a systematic literature search strategy; consistent results with sufficient numbers of well-designed studies; criteria-based evaluation of overall scientific strength and quality of included studies and definitive conclusions; national expertise clearly evident; developed or revised within the past five years.

#### **B** Good quality

Material officially sponsored by a professional, public, or private organization or a government agency; reasonably thorough and appropriate systematic literature search strategy; reasonably consistent results, sufficient numbers of well-designed studies; evaluation of strengths and limitations of included studies with fairly definitive conclusions; national expertise clearly evident; developed or revised within the past five years.

#### C Low quality or major flaw

Material not sponsored by an official organization or agency; undefined, poorly defined, or limited literature search strategy; no evaluation of strengths and limitations of included studies; insufficient evidence with inconsistent results; conclusions cannot be drawn; not revised within the past five years.

#### Quality Rating for Organizational Experience (Level V)

#### A High quality

Clear aims and objectives; consistent results across multiple settings; formal quality improvement or financial evaluation methods used; definitive conclusions; consistent recommendations with thorough reference to scientific evidence.

#### **B** Good quality

Clear aims and objectives; formal quality improvement or financial evaluation methods used; consistent results in a single setting; reasonably consistent recommendations with some reference to scientific evidence.

#### C Low quality or major flaws

Unclear or missing aims and objectives; inconsistent results; poorly defined quality; improvement/financial analysis method; recommendations cannot be made.

Quality Rating for Case Report, Integrative Review, Literature Review, Expert Opinion, Community Standard, Clinician Experience, Consumer Preference (Level V)

#### A High quality

Expertise is clearly evident, draws definitive conclusions, and provides scientific rationale; thought leader in the field.

#### **B** Good quality

Expertise appears to be credible, draws fairly definitive conclusions, and provides logical argument for opinions.

#### C Low quality or major flaws

Expertise is not discernable or is dubious; conclusions cannot be drawn.

#### 2017 Appendix G Individual Evidence Tool

Appendix G Individual Evidence Summary Tool

| | EBP Question: | | | | | |
|---|---|---|---|---|---|---|
| Article Author and Date | | Sample, Sample<br>Size, Setting | Findings That Help<br>Answer the EBP<br>Question | Observable<br>Measures | Limitations | Evidence Level,<br>Quality |
| | | D N/A | | | | |
| | | D N/A | | | | |
| | | □ N/A | | | | |
| | | □ N/A | | | | |
| | | □ N/A | | | | |
| | | □ N/A | | | | |
| | | □ N/A | | | | |
| | Author and Date | | Size, Setting I N/A I N/A | Author and Date Evidence Type Sample, Sample Size, Setting Findings That Help Answer the EBP Question N/A N/A N/A | Author and Date Evidence Type Sample, Sample Answer the EBP Question Observable Measures ON/A N/A N/A | Author and Date Evidence Type Sample, Sample Size, Setting Findings That Help Answer the EBP Question Umitations I N/A I N/A I N/A I N/A I N/A |

Attach a reference list with full citations of articles reviewed for this EBP question.

#### Directions for Use of the Individual Evidence Summary Tool

#### **Purpose**

This form is used to document the results of evidence appraisal in preparation for evidence synthesis. The form provides the EBP team with documentation of the sources of evidence used, the year the evidence was published or otherwise communicated, the information gathered from each evidence source that helps the team answer the EBP question, and the level and quality of each source of evidence.

#### **Article Number**

Assign a number to each reviewed source of evidence. This organizes the individual evidence summary and provides an easy way to reference articles.

#### **Author and Date**

Indicate the last name of the first author or the evidence source and the publication/communication date. List both author/evidence source and date.

#### **Evidence Type**

Indicate the type of evidence reviewed (e.g., RCT, meta-analysis, mixed methods, qualitative, systematic review, case study, narrative literature review).

#### Sample, Sample Size, and Setting

Provide a quick view of the population, number of participants, and study location.

#### Findings That Help Answer the EBP Question

Although the reviewer may find many points of interest, list only findings that directly apply to the EBP question.

#### **Observable Measures**

QuaNtitative measures or variables are used to answer a research question, test a hypothesis, describe characteristics, or determine the effect, impact, or influence. QuaLitative evidence uses cases, context, opinions, experiences, and thoughts to represent the phenomenon of study.

#### Limitations

Include information that may or may not be within the text of the article regarding drawbacks of the piece of evidence. The evidence may list limitations, or it may be evident to you, as you review the evidence, that an important point is missed or the sample does not apply to the population of interest.

#### **Evidence Level and Quality**

Using information from the individual appraisal tools, transfer the evidence level and quality rating into this column.

#### 2017 Appendix H Evidence Synthesis and Recommendation Tool



#### **Key Points:**

- Evidence synthesis is best done through group discussion. All team members share their perspectives, and the team uses critical thinking to arrive at a judgment based on consensus during the synthesis process. The synthesis process involves both subjective and objective reasoning by the full EBP team. Through reasoning, the team:
  - Reviews the quality appraisal of the individual pieces of evidence
  - Assesses and assimilates consistencies in findings
  - Evaluates the meaning and relevance of the findings
  - Merges findings that may either enhance the team's knowledge or generate new insights, perspectives, and understandings
  - Highlights inconsistencies in findings
  - Makes recommendations based on the synthesis process
- When evidence includes multiple studies of Level I and Level II evidence, there is a similar population or setting of interest, and there is consistency across findings, EBP teams can have greater confidence in recommending a practice change. However, with a majority of Level II and Level III evidence, the team should proceed cautiously in making practice changes. In this instance, recommendation(s) typically include completing a pilot before deciding to implement a full-scale change.
- Generally, practice changes are not made on Level IV or Level V evidence alone. Nonetheless, teams have a variety of options for actions that include, but are not limited to: creating awareness campaigns, conducting informational and educational updates, monitoring evidence sources for new information, and designing research studies.
- The quality rating (see Appendix D) is used to appraise both individual quality of evidence and overall quality of evidence.

#### Appendix H

5ynthesis Process and Recommendations Tool

| EBP Question: | | | |
|---|---|---|---|
| Category (Level Type) | Total Number of<br>Sources/Level | Overall Quality<br>Rating | Synthesis of Findings<br>Evidence That Answers the EBP Question |
| Level I | | | |
| Epperimental study Izandomized controlled Mal (RCT) Systematic review of RCTs with or without meta-analysis Epplanatory mixed method design that includes only a teret I qualititative study | | | |
| Level II | | | |
| <ul> <li>Quasi-experimental studies</li> <li>Systematic review of a combination of RCTs and quasi-experimental studies, or quasi-experimental studies only, with or without meta-analysis</li> <li>Explanatory mixed method design that includes only a Level II quaNtitative study</li> </ul> | | | |
| Level III | | | |
| <ul> <li>Nonexperimental study</li> <li>Systematic review of a combination of RCTs, quasi-experimental and nonexperimental studies, or nonexperimental studies only, with or without meta- analysis</li> <li>Qualitative study or meta- synthesis</li> <li>Exploratory, convergent, or multiphasic mixed-methods studies</li> <li>Explanatory mixed method design that includes only a level III Qualtitative study</li> </ul> | | | |

@2017 The Johns Hopkins Hospital/ The Johns Hopkins Universit

#### Appendix H

Synthesis Process and Recommendations Tool

| + | | | | |
|---|---|---|---|---|
| | Category (Level Type) | Total Number of<br>Sources/Level | Overall Quality<br>Rating | Synthesis of Findings<br>Evidence That Answers the EBP Question |
| | Level IV | | | |
| | <ul> <li>Opinions of respected authorities and/or<br/>reports of nationally recognized expert<br/>committees or consensus panels based on<br/>scientific evidence</li> </ul> | | | |
| ľ | Level V | | | |
| | <ul> <li>Evidence obtained from literature or<br/>integrative reviews, quality improvement,<br/>program evaluation, financial evaluation, or<br/>case reports</li> </ul> | | | |
| | <ul> <li>Opinion of nationally recognized expert(s)</li> <li>based on experiential evidence</li> </ul> | | | |

Based on your synthesis, which of the following four pathways to translation represents the overall strength of the evidence?

- □ **Strong, compelling evidence, consistent results**: Solid indication for a practice change is indicated.
- □ **Good and consistent evidence**: Consider pilot of change or further investigation.
- □ **Good but conflicting evidence**: No indication for practice change; consider further investigation for new evidence or develop a research study.
- □ **Little or no evidence**: No indication for practice change; consider further investigation for new evidence, develop a research study, or discontinue project.

If you selected either the first option or the second option, **continue**. If not, **STOP**, translation is not indicated.

Recommendations based on evidence synthesis and selected translation pathway

#### Consider the following as you examine fit:

#### Are the recommendations:

- Compatible with the unit/departmental/organizational cultural values or norms?
- Consistent with unit/departmental/organizational assumptions, structures, attitudes, beliefs, and/or practices?
- Consistent with the unit/departmental/organizational priorities?

#### Consider the following as you examine feasibility:

- Can we do what they did in our work environment?
- Are the following supports available?
  - Resources
  - Funding
  - Approval from administration and clinical leaders
  - Stakeholder support
  - Is it likely that the recommendations can be implemented within the unit/department/organization?

#### **Directions for Use of This Form**

#### Purpose of form

Use this form to compile the results of the individual evidence appraisal to answer the EBP question. The pertinent findings for each level of evidence are synthesized, and a quality rating is assigned to each level.

#### Total number of sources per level

Record the number of sources of evidence for each level.

#### Overall quality rating

Summarize the overall quality of evidence for each level. Use Appendix D to rate the quality of evidence.

#### Synthesis of findings: evidence that answers the EBP question

- Include only findings from evidence of A or B quality.
- Include only statements that directly answer the EBP question.
- Summarize findings within each level of evidence.
- Record article number(s) from individual evidence summary in parentheses next to each statement so that the source of the finding is easy to identify.

# Develop recommendations based on evidence synthesis and the selected translation pathway

Review the synthesis of findings and determine which of the following four pathways to translation represents the overall strength of the evidence:

- Strong, compelling evidence, consistent results: Solid indication for a practice change.
- Good and consistent evidence: Consider pilot of change or further investigation.
- Good but conflicting evidence: No indication for practice change; consider further investigation for new evidence or develop a research study.
- Little or no evidence: No indication for practice change; consider further investigation for new evidence, develop a research study, or discontinue the project.

#### Fit and feasibility

Even when evidence is strong and of high quality, it may not be appropriate to implement a change in practice. It is crucial to examine feasibility that considers the resources available, the readiness for change, and the balance between risk and benefit. Fit refers to the compatibility of the proposed change with the organization's mission, goals, objectives, and priorities. A change that does not fit within the organizational priorities will be less likely to receive leadership and financial support, making success difficult. Implementing processes with a low likelihood of success wastes valuable time and resources on efforts that produce negligible benefits.

# 2017 Appendix I Action Planning Tool

| 1. Complete the following activities to ensure successful translation: | | |
|---|---|---|
| □ Secure a project leader. | | |
| □ Identify change champions. | | |
| <ul> <li>Consider whether translation</li> </ul> | □ Consider whether translation activities require different or additional members. | |
| □ Schedule time to complete n | □ Schedule time to complete milestones. | |
| <ul> <li>Identify critical milestones ar</li> </ul> | nd related tasks. | |
| □ Identify observable pre or po | ost measures. | |
| 2. Identify barriers to the success of the change, and then identify strengths that can be leveraged to overcome barriers. | | |
| Barriers | Resources or Strengths | Plan to Overcome Barriers by Leveraging Strengths as Appropriate |
| 3. Consider whether or how this change will affect the following: | | |
| ☐ Electronic health record | ☐ Workflow | ☐ Policies and/or procedures |
| 4. Confirm support and/or availability of funds to cover expenses. (Check all that apply) | | |
| <ul><li>Personnel costs</li></ul> | ☐ Educ | ☐ Education or further training |
| □ Supplies/equipm | nent | ☐ Content or external experts |
| □ Technology | ☐ Disse | emination costs (conference costs, |
| <ul><li>Photocopying</li></ul> | trave | · |
| ., 0 | □ Othe | □ Other: |

| | 5. Identify critical milestones and related tasks: |
|---|---|
| | (Insert Milestone 1) (Insert Milestone 2) (Insert Milestone 3) (Insert Milestone 3) |
| | (languat to als) |
| | (Insert task) |
| Tasks | |
| Ta | |

## **Directions for Use of the Action Planning Tool**

#### **Purpose of form**

This form is used to guide you as you create an action plan.

#### Activities to ensure successful translation

These are all activities that must be completed as you plan the change. Consider pre- and post-observable measures that can be used to determine whether the change was successful. In addition, identifying critical milestones allows the team to see whether they are on track to accomplish the goals.

# Identify strengths/resources and barriers to the success of the change

This analysis allows teams to identify barriers to implementation and potentially mitigate them using inherent strengths and resources. You may find specific challenges that will likely impact the ability to deliver on the action plan. Though these obstacles can get in the way, knowing about them up front is helpful so that you can engage support and create a plan to address them.

# Consider whether or how the change will impact workflows and processes

Be mindful of the impact of the change downstream. For example, will changes need to be made to the electronic medical record to accommodate the change, or will this change impact the workflow of any other staff who have not been considered?

#### Confirm support and/or availability of funds to cover expenses

Use this as a guide to prompt thoughtfulness about financial obligations that may be a part of the rollout.

#### Identify critical milestones and related tasks

Consider all the categories of work (milestones) necessary to implement this change. What tasks must be accomplished first for each milestone in order to move forward? When must they be completed to stay on track? For example, if a milestone is to implement a protocol, list all tasks to accomplish it.

# 2017 Appendix J Dissemination Tool

| 1. Think about the project findings and practice change initiative. What is the most important information you need to convey? | | |
|---|---|---|
| 2. Align key messages with audiences. | | |
| Audience | Key Message | Communication Method |
| Interdisciplinary stakeholders | | |
| Organizational leadership | | |
| Departmental leadership | | |
| Frontline staff | | |
| External community (publications, posters, and presentations) | | |
| 3. Review examples below to | o identify appropriate communicat | tion methods. |
| <ul> <li>Written publication</li> <li>Online program</li> <li>External conference</li> <li>Podium presentation</li> <li>Poster presentation</li> <li>Social media blast</li> <li>Internal meeting/inservice</li> <li>Audio/video content</li> <li>Others:</li> </ul> | | |

#### **Directions for Use of the Dissemination Tool**

#### **Purpose**

This form is useful at various points in the EBP project process. It is usually completed toward the end of the project, when findings are known and efforts have produced a product, tool, program, or policy.

#### Align key message with audience

Think about the project findings. What has the project effort accomplished? What products, policy changes, or outcomes can you report? Identify the end users—who is your audience? Your audience may be individuals, organizations, or networks who might have an interest in the project outcomes.

#### **Communication method**

This is the communication plan, and it can occur on many levels. Think about reaching the varied audiences using a multitude of methods. These can include, but are not limited to, written text, audio / visual content, online programs, and poster presentations.

#### **ANNEX 2:**

# Clinical Effectiveness and Evidence Based Practice Questionnaire (EBPQ).

This questionnaire is designed to gather information and opinions on the use of evidence based practice amongst health professionals. There are no right or wrong answers for we are interested in *your* opinions and *your* own use of evidence in *your* practice.

- 1) Considering your practice in relation to an individual patient's care over the past year, how often have you done the following in response to a gap in your knowledge (please V or X):
- a) Formulated a clearly answerable question as the beginning of the process towards filling this gap:

 ?
 ?
 ?
 ?
 ?
 ?
 ?
 ?
 1
 1
 2
 3
 4
 5
 6
 7
 5
 7
 6
 Never
 Frequently

b) Tracked down the relevant evidence once you have formulated the question

 ?
 ?
 ?
 ?
 ?
 ?
 ?
 ?
 ?
 1
 1
 2
 3
 4
 5
 6
 7
 7
 7
 Never
 Frequently

c) Critically appraised, against set criteria, any literature you have discovered

 ?
 ?
 ?
 ?
 ?
 ?
 ?
 ?
 1
 1
 2
 3
 4
 4
 5
 6
 7
 Frequently

| ?<br>1<br>Never<br>e) | ②<br>2<br>Evaluated the out | ?<br>3<br>come | s of yo | ū<br>z<br>our pra | 1 | | ?<br>5 | | ?<br>6 | ?<br>7<br>Frequently |
|---|---|---|---|---|---|---|---|---|---|---|
| ?<br>1<br>Never | ?<br>2 | ? | | [ | | | ?<br>5 | | ?<br>6 | ⑦<br>7<br>Frequently |
| f) 1 Never | Shared this inform 2 2 Please indicate ( of the following | ?<br>3<br>by √ ( | or X) v | where | on th | e scal | ②<br>5 | would | 2<br>6<br>I place yourse | 7<br>Frequently<br>If for each |
| My workload is too great<br>for me to keep up to date<br>with all the new evidence | | | | | | | _ | | New evidence important the time in machedule | at I make<br>ny work |
| practice o | aving my clinical<br>luestioned<br>based practice is<br>f time | | | | | | | | I welcome que on my practice Evidence base practice is fundamental professional pro | ed<br>to |
| methods | ried and trusted<br>rather than<br>to anything new | | | | | | | | My practice has changed because of evidence I have found | |

d) Integrated the evidence you have found with your expertise:
## 3) On a scale of 1 to 7 (with 7 being the best) how would you rate your

| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
|---|---|---|---|---|---|---|---|
| Research skills | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| IT skills | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Monitoring and reviewing of practice skills | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Converting your information needs into a research question | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Awareness of major information types and sources | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Ability to identify gaps in your professional practice | Poor | | | | | | Best |
| · | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Knowledge of how to retrieve evidence | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Ability to analyse critically evidence against set standards | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Ability to determine how valid (close to the truth) the material is | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Ability to determine how useful (clinically applicable) the material is | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Ability to apply information to individual cases | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Sharing of ideas and information with colleagues | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Dissemination of new ideas about care to colleagues | Poor | | | | | | Best |
| | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| Ability to review your own practice | Poor | | | | | | Best |

## 4) Finally, some information about you:

Your profession: Year qualified:

Your position/grade: Your speciality:

## Please circle the most appropriate answer as it concerns you:

Your sex: Male Female

Your age range: 20-29 30-39 40-49 50-59 60-69

## **ANNEX 3:**

## **Managers' Consent Form**



## TERMO DE ANUÊNCIA DOS GESTORES DE ÁREA

PESQUISADOR RESPONSÁVEL: Profª Drª Eliseth Ribeiro Leão

TÍTULO DO PROJETO: Pratica Baseada em Evidências: Proposta de Aplicação de Ferramentas Facilitadoras para os Enfermeiros Clínicos.

VIGÊNCIA: 01.12.2019 a 01.03.2021

Nós, abaixo assinados, declaramos ser de nosso conhecimento o teor do projeto acima, cujos participantes têm a nossa anuência em desenvolver as atiylidades descritas no projeto proposto,

pertinentes à nossa área de gestão.

Nome do gestor da área solicitante Setor: Faculdade Israelita de Ciência da Saúde Albert Einstein

Data: 11. 11. 2019

Claudia Regina Laselva
Claudia Regina Laselva
Claudia Regina Albert Einstein
Directora Unidade Hospital Israelita Albert Einstein

Prof<sup>a</sup> Dra. Andréa Gomes da Costa Mohallem Vice-Diretora Faculdade Israelita de Ciências da Saúde Albert Einstein

Nome do gestor da área de realização

CLAUDIA REGINA LASSELVI

Setor: Diretoria Assistencial Hospital Albert Einstein

Data: 11.11.2019

Assinatura Carimbo

## Annex 4:

## **Researcher's Term of Commitment**

## TERMO DE COMPROMISSO DO PESQUISADOR RESPONSÁVEL

Eu, Profª Dra Eliseth Ribeiro Leão, pesquisador responsável do Projeto intitulado Pratica Baseada em Evidências: Proposta de Aplicação de Ferramentas Facilitadoras para os Enfermeiros Clínicos, declaro estar ciente do compromisso de manter as informações pertinentes a esse projeto atualizadas no Sistema de Gerenciamento de Projetos de Pesquisa (SGPP), incluindo a entrega dos relatórios científicos, apresentando as entregas propostas no projeto (artigo, melhoria de processo ou formação acadêmica). Estou também ciente de que, no caso de tecnologia passível de proteção industrial (patentes ou modelos de utilidade) resultante do projeto em questão e, antes da divulgação oral e/ou escrita da pesquisa realizada, deverei comunicar o conteúdo da mesma ao Centro de Inovação Tecnológica (CIT). Por fim, declaro estar ciente das diretrizes de Boas Práticas Científicas, bem como me comprometo a seguir os códigos de ética em pesquisa e de integridade científica (http://web.telaviva/home/portal-de-pesquisa/fazendo-pesquisa-com-etica/fazendo-pesquisa-com-etica.html)

São Paulo, 11 de novimbro, 2019

ELiseth Ripoiro LEAD

Nome do pesquisador responsável do Projeto

**Assinatura** 

## Annex 5:

## **Participants' Term of Consent**



#### TERMO DE ANUÊNCIA DOS PARTICIPANTES DE PROJETO

PESQUISADOR RESPONSÁVEL: Profª Drª Eliseth Ribeiro Leão

TÍTULO DO PROJETO: Pratica Baseada em Evidências: Proposta de Aplicação de Ferramentas Facilitadoras para os Enfermeiros Clínicos.

VIGÊNCIA: 01.12.2019 a 01.03.2021

Nós, abaixo assinados, declaramos a nossa anuência em participar deste projeto e de estar cientes das obrigações constantes do regulamento do SGPP e das diretrizes de Boas Práticas Científicas, bem como nos comprometemos a seguir os códigos de ética em pesquisa e de integridade

| científica. | /: |
|---|---|
| Eliseth RiBeiro LEAD | The state of the s |
| Nome do participante do Projeto<br>Instituição/Departamento<br>Liduale Staves Jackeda Conta | Assinatura Corta |
| Nome do participante do Projeto<br>Instituição/Departamento | Assinatura |
| Nome do participante do Projeto<br>Instituição/Departamento | Assinatura |

São Paulo, OI de Norkmho \_\_\_\_, 20\_19

## **APPENDICES**

## **Appendix 1:** Authorization document for translating the Johns Hopkins Center for Evidence-Based Practice tools



Kim



Kim Bissett, MSN, MBA, RN Nurse Educator, EBP Specialist Institute for Johns Hopkins Nursing

## Appendix 2:

# QUESTIONNAIRE TO CHECK THE SUITABILITY OF THE AUTHORIZED TRANSLATION OF THE PORTUGUESE LANGUAGE VERSION OF THE JOHNS HOPKINS PBE GUIDE TOOLS

## Sociodemographic data

| Expert name: |
|---|
| Length of experience in Evidence-based practice: |
| Highest academic level: |
| Occupation area: |
| Check the answer that most closely matches your assessment regarding the tradition of the content of the following tools: |
| APPENDIX A: PET Management Guide |
| APPENDIX B: Development of the question |
| APPENDIX C: Stakeholder analysis |
| APPENDIX D: Evidence and quality level guide |
| APPENDIX E: Research Evidence Assessment Tool |
| APPENDIX F: Non-Research Evidence Assessment Tool |
| APPENDIX G: Individual Evidence Tool |
| APPENDIX H: Evidence and Recommendations Synthesis Tool |
| APPENDIX I: Action Planning Tool |

APPENDIX J: Dissemination Tool

| 1)Are the translations intelligible? | | | | |
|---|---|---|---|---|
| | ( | )YES | ( | )NO |
| 2)Are | th | ere any sugge | sti | ons for changes? |
| | ( | )YES | ( | )NO |
| 3)If y | es, | | | |

| Which tool | Which change |
|------------|--------------|

## Appendix 3:

## PBE guiding tools for the Johns Hopkins Nursing Evidence-based Practice (versions translated into Portuguese)

Apêndice A - PET Guia de Gerenciamento

Apêndice B - Desenvolvimento da Pergunta

Apêndice C - Análise de Partes Interessadas

Apêndice D - Guia de Nível de Evidência e Qualidade

Apêndice E - Ferramenta de Avaliação de Evidência de Pesquisa

Apêndice F - Ferramenta de Avaliação de Evidências que não sejam de Pesquisa

Apêndice G - Ferramenta de Evidência Individual

Apêndice H - Ferramenta de Síntese de Evidências e Recomendações

Apêndice I - Ferramenta de Planejamento de Ações

Apêndice J - Ferramenta de Disseminação

## Apêndice A - PET Guia de Gerenciamento



## Pergunta Prática

- Passo 1: Recrutar equipe multiprofissional
  - Passo 2: Definir o problema
  - Passo 3: Desenvolver e refinar a questão de PBE
  - Passo 4: Identificar as partes interessadas
  - Passo 5: Determinar a responsabilidade da liderança do projeto
  - Passo 6: Agendar reuniões da equipe

## **Evidência**

- Passo 7: Realizar buscas internas e externas por evidências
- Passo 8: Avaliar o nível e a qualidade de cada evidência
- Passo 9: Resumir individualmente a evidência
- Passo 10: Sintetizar a força geral e a qualidade da evidência
- Passo 11: Desenvolver recomendações para mudanças baseadas na síntese de evidências
  - Evidência forte e convincente, resultados consistentes.
  - Boa evidência, resultados consistentes
  - Boa evidência, resultados conflitantes
  - Evidência insuficiente ou ausente

## Tradução

Passo 12: Determinar ajustes, viabilidade e adequação das recomendações para implementação / tradução.

Passo 13: Cria plano de ação

Passo 14: Garantir apoio e recursos para implementar plano de ação

Passo 15: Implementar plano de ação

Passo 16: Avaliar resultados

Passo 17: Relatar resultados para as partes interessadas

Passo 18: Identificar os próximos passos

Passo 19: Divulgar os achados

| Data<br>Início | Dias<br>Requeridos | Data<br>Final | Respon-<br>sável | Marco<br>Histórico | Comentários /<br>Recursos<br>Necessários |
|---|---|---|---|---|---|
| | | | | - | |

## Apêndice B - Desenvolvimento da Pergunta

| 1. Qual é o problema? | |
|---|---|
| 2. Porque o problema é importante ou relevante | ? O que aconteceria se não fosse abordado? |
| 3. Qual é a prática atual? | |
| 4. Como o problema foi identificado? (Marque t | odos os itens que se aplicam) |
| <ul> <li>Questões de segurança e gestão de riscos</li> </ul> | □ Variações da prática com o preconizado |
| <ul> <li>Preocupações com a qualidade (eficiência, eficácia,<br/>oportunidade, equidade, centralização no paciente)</li> </ul> | <ul> <li>Variações da prática comparado aos padrões da<br/>comunidade</li> </ul> |
| ☐ Insatisfação do paciente, colaboradores ou | □ Prática atual não validada |
| resultados organizacionais | □ Preocupações financeiras |
| 5. Quais são os componentes do PICO? | |
| <b>P</b> – (Paciente, população, ou problema) | |
| I – (Intervenção) | |
| C – (Comparação com outras intervenções, se neces | sário) |
| <ul> <li>O – (Resultados: Os resultados são medidas qualit<br/>da mudança)</li> </ul> | rativas ou quantitativas para determinar o sucesso |
| | ica 🛚 Questão Clínica |

| 7. Listar possiveis descritores, base de dados para pesquisa e estrategias de pesquisa. | | | | | |
|---|---|---|---|---|---|
| 8. Quais evidê | ncias devem ser | coletadas? (Mar | que todos os ite | ns que se aplica | m) |
| □ Publicações | (e.g., PubMed, M | EDLINE, LILACS, | Cochrane, etc) | | |
| □ Padrões (reg | gulatórios, profissi | onais, comunitário | os) | | |
| <ul><li>Diretrizes</li></ul> | | | | | |
| <ul><li>Dados orgar família)</li></ul> | nizacionais (e.g., d | lados financeiros, | experiência clínic | a local, preferênci | as do paciente e |
| □ Declaração | de posicionamento | o | | | |
| 9. Pergunta cli | nica de PBE revi | sada | | | |
| revisão pode | estar na formulaçã | odem não ser evido<br>ão da questão básio<br>ara questão clínica | ca (background qu | estion) ou até nas l | |
| 10. Plano de m | edeição dos resi | ultados | | | |
| O que vamos<br>medir?<br>(Estrutura,<br>processo,<br>resultado) | Como vamos<br>medir isso?<br>(métricas<br>expressas como<br>taxas ou<br>porcentagens) | Qual será a<br>periodicidade da<br>medição?<br>(frequência) | Onde vamos<br>obter os<br>dados? | Quem coletará<br>os dados? | Para quem<br>vamos relatar os<br>dados? |
| por some gone, | | | | | |

## Instruções para o uso da Ferramenta de Desenvolvimento da Pergunta Clínica

## Objetivo

Este formulário é utilizado para Desenvolvimento de pergunta de PBE, guia a equipe no processo de busca de evidências. A pergunta, os descritores, a estratégia de pesquisa e as fontes de evidencias podem ser revisadas à medida que a equipe de PBE refina a pergunta de PBE.

## Qual é o problema e porque ele é importante?

Indique porque o projeto foi realizado. O que levou a equipe a buscar evidências? Certifique-se que a formulação do problema defina o problema atual e não inclua uma solução. Sempre que possível quantifique a extensão do problema e valide a descrição final do problema com a equipe envolvida na prática. É importante que a equipe multiprofissional dedique tempo em grupo para refletir, reunir informações, observar a prática atual, ouvir o corpo clínico, visualizar como o processo poder ser diferente ou melhorado, sondar e analisar a descrição do problema de modo que desenvolva uma compreensão compartilhada da equipe com a descrição do problema.

## Qual é a prática atual?

Defina a prática atual no que se refere ao problema. Reflita sobre as políticas e procedimentos atuais, observe as práticas. O que você vislumbra?

## Como o problema foi identificado?

Verifique todas as descrições que se aplicam.

## Quais são os componentes do PICO?

- P (Paciente, população, problema) Por exemplo: idade, sexo, cenário, etnia, condição, doença, tipo de paciente ou população.
- I (Intervenção) Por exemplo: tratamento, medicação, educação, exames diagnósticos ou melhores práticas.
- **C** (Comparação com outras intervenções ou prática atual para questões clínicas (Foreground questions), não é aplicável para questões básicas (Background questions) que identificam as melhores práticas).
- **O** (Resultados) Descritos em termos mensuráveis, pode ser uma estrutura, um processo ou uma medida de resultado com base na mudança desejada (por exemplo: diminuição de quedas, diminuição no tempo de hospitalização, aumento na satisfação do paciente.

## Pergunta Inicial de PBE

Uma pergunta inicial (geralmente uma pergunta básica [background question] que é frequentemente refinada e ajustada à medida que a equipe realiza a pesquisa na literatura):

- Perguntas Básicas (Background questions) são amplas e adotadas quando a equipe tem pouco conhecimento ou experiência na área de interesse. As perguntas básicas são utilizadas geralmente para identificar as melhores práticas.
- Perguntas Clínicas (Foreground questions) são focadas, com comparações específicas de duas ou mais ideias ou intervenções. Perguntas clínicas fornecem um conjunto (corpo) específico relacionado à pergunta de PBE. As perguntas clínicas geralmente fluem da pergunta básica somada à revisão da literatura.

## Lista de possíveis descritores, base de dados para pesquisa e estratégias de pesquisa

Usando os componentes do PICO e a pergunta inicial de PBE, liste os descritores. Os descritores podem ser adicionados ou ajustados por meio da pesquisa de evidências. Documente os descritores, a estratégia de pesquisa e os bancos de base de dados consultados com detalhes suficientes para replicação.

## Quais evidências devem ser coletadas?

Verifique os tipos de evidências que a equipe coletará com base no PICO e na pergunta inicial de PBE.

## Pergunta de PBE revisada

Muitas vezes a pergunta que você começa pode não ser a pergunta final de PBE. Perguntas básicas podem ser refinadas e modificadas para perguntas clínicas baseado na revisão de evidências. As perguntas clínicas são perguntas focalizadas que incluem comparações específicas e produzem uma faixa de evidência mais restrita.

#### Plano de mensuração

As mensurações podem ser adicionadas ou modificadas à medida que a revisão da literatura é completada, iniciando o planejamento da tradução:

- Uma medida é uma quantidade ou um grau de algo, como por exemplo, número de quedas com dano. Cada medida deve ser convertida em uma métrica, que deve ser calculada antes e depois da implementação da alteração.
- As métricas permitem que você saiba se a mudança foi bem sucedida. Possuem um numerador e um denominador e são normalmente expressos como taxas ou porcentagens. Um exemplo de métrica quanto ao número de quedas com dano (numerador) dividido por 1.000 pacientes-dia (denominador). Outros exemplos de métricas incluem o número de RNs que recebem assistência direta (numerador) dividido pelo número de funcionários que prestam assistência direta, ou o número de erros de medicações dividido por 1.000 prescrições.

## Apêndice C - Análise de Partes Interessadas

| 1. | Identifique os | principais interessados | | | |
|---|---|---|---|---|---|
| | Gerente ou coordenador direto | | | □ Líderes organizacio | onais |
| | _ ` . | | <ul> <li>Membros da equipe multidisciplinar (por exemplo:<br/>médicos, nutricionistas, fisioterapeutas, terapeuta</li> </ul> | | |
| | | | | medicos, nutricionis ocupacional) | stas, fisioterapeutas, terapeuta |
| | Pacientes e / pacientes e fa | ou famílias, comitê consultivo o<br>amiliares. | de | <ul><li>□ Administradores</li><li>□ Outras unidades ou departamentos</li><li>□ Outros:</li></ul> | |
| | Organizações | profissionais | | | |
| ۵ | Comitês | | | | |
| (A: | s funções das pa | sponsabilidades dos principa<br>artes interessadas incluem: respon<br>correspondentes estão descritas | nsab | ilidade, consulta, aprovaç | |
| Responsabilidade • Identificar tarefas completas • Recomendar uma autoridade | | | Co | <ul><li>Fornece contribuiç<br/>assunto)</li><li>Sem autoridade de</li></ul> | ões (por ex. especialistas no ecisória |
| Aprovação | | Inf | <ul><li>Informação</li><li>Notificação de progresso e mudanças</li><li>Sem contribuições decisórias</li></ul> | | |
| Γaι | refas do | Nome do interessado | Nome do interessado | | Nome do interessado |
| Pro | ojeto | Função do interessado | Função do interessado | | Função do interessado |

## Instruções para uso da Ferramenta de Análise das partes interessadas

Este formulário é utilizado para identificar os principais interessados. Esse são pessoas, grupos ou departamentos da organização que têm interesse ou preocupação com seu projeto e / ou podem ajuda-lo a garantir recursos para implementar seu plano de ação. Envolva as partes interessadas no início do seu processo para garantir adesão.

## Definição

Os Stakeholders são "pessoas ou grupos que possuem interesse em uma decisão clínica [ou não clínica] e nas evidências que apoiam essa decisão" (AHRQ, 2014).

## Identifique os principais interessados

Identifique os 5-7 principais interessados que mais podem afetar, ou quem serão mais afetados pelo projeto, ações, objetivos ou mudanças e quem pode influenciar no sucesso do trabalho de tradução. Os principais "stakeholders" são indivíduos ou grupos que:

- Tomam decisões sobre o projeto
- · Aprovam o projeto ou aspectos do projeto
- Servem como especialista no assunto
- Fornecem recursos como: suporte, mudanças em políticas, recursos e tempo.

## Análise das partes interessadas

É útil considerar quais dos quarto papéis que cada parte interessada pode desempenhar no seu planejamento de ação e trabalho de tradução. As possíveis funções são:

- Responsabilidade
- Aprovação
- Consulta
- Informação

Lembre-se de que uma parte interessada pode preencher papéis diferentes, dependendo da ação. A conclusão da ferramenta de análise das partes interessadas ajudará a esclarecer papéis e responsabilidades. As descrições de responsabilidades para cada função fornecida no formulário serão úteis nesse processo.

Referências: Agency for Healthcare Research and Quality. (2014) .Stakeholder Guide 2014. Retrieved from www.effectivehealthcare.ahrq.gov.AHRQ Publication No. 14-EHC010-EF. Replaces Publication No. 11-EHC069-EF

## Apêndice D - Guia de Nível de Evidência e Qualidade

## Apêndice D

Níveis de Evidência

Nível de Evidencia e Guia de Qualidade

| Nível I | Estudos Quantitativos |
|---|---|
| Estudo experimental, ensaio clínico<br>randomizado (RCT). | A <u>Alta qualidade</u> : Resultados consistentes e generalizáveis, tamanho de amostra suficiente para o desenho do estudo, controle adequado, conclusões definitivas. Recomendações consistentes baseado em revisões abrangentes da literatura que incluam referências comidetas a evidência científica. |
| Desenho de método misto explanatório, que<br>inclui apenas um estudo quantitativo de Nível<br>I. | B <u>Boa qualidade</u> : Resultados razoavelmente consistentes, tamanho de amostra suficiente para o desenho do estudo, algum controle, conclusões bastante definitivas. Recomendações razoavelmente consistentes baseadas em revisão da literatura razoavelmente abrangentes que inclua alguma referência a evidências científicas. |
| Revisão sistemática de <u>RCTs</u> , com ou sem<br>meta-análise. | C <u>Baixa qualidade ou grandes falhas</u> : Pouca evidência e com resultados inconsistentes, tamanho insuficiente da amostra para o tamanho do estudo, conclusões não podem ser <u>deligradas</u> |
| Nível II | Estudos Qualitativos |
| Estudo quase-experimental. | |
| Desenho de método misto explanatório, que<br>inloui, apenas um estudo quantitativo de Nível<br>II. | Não existem princípios comumente acordados para julgar a qualidade dos estudos qualitativos. É um processo subjetivo baseado na extensão em que os dados do estudo contribuem para a síntese e quanta informação é conhecida sobre os esforços dos pesquisadores para atender aos critérios de avaliação. |
| Revisão sistemática de uma combinação de<br>RCTs, e estudos quase-experimentais, ou<br>somente estudos quase-experimentais, com | Para meta-sínteses, há concordância preliminar de que avaliações de qualidade individual dos estudos devem ser feitas antes da síntese para excluir estudos de beixa qualidade. A/B Alta/Boa qualidade é utilizada para estudos únicos e meta-sínteses². |
| ou sem meta-análise . | |
| Nível III<br>Estudo não:experimental. | O relatório discute os esforços para melhorar ou avaliar a qualidade e a investigação garal com detalhes suficientes,<br>descreve as técnicas específicas usadas para melhorar a qualidade da pesquisa. Evidência de alguns ou todos os itens<br>a seguir são encontrados no relatório: |
| Revisão sistemática de uma combinação de | <ul> <li>Transperência: Descrevem como as informações foram documentadas para justificar decisões, como os dados<br/>foram revisados por outras pessoas e como os temas e categorias foram formuladas.</li> </ul> |
| RCTs, estudos quase-experimentais e não-<br>experimentais, ou estudos não experimentais | <ul> <li>Diligência: Ler e reler os dados para checar interpretações, buscar oportunidades para buscar múltiplas fontes<br/>para corroborar exidencias.</li> </ul> |
| apenas, com ou sem meta-análise. | <ul> <li>Verificação: O processo de verificação, confirmação, e garantia de coerência metodológica.</li> </ul> |
| Estudos de métodos mistos exploratórios,<br>convergentes ou multifásicos. | <ul> <li>Auto-reflexão e escrutínio: Estar continuamente consciente de como as experiências, antecedentes ou<br/>preconceitos de um pesquisador pode moidar e influenciar análises e interpretações.</li> </ul> |
| Desenho de método misto explanatório, que | <ul> <li>Pesquisa orientada por participantes: Os participantes moldam o escopo e a abrangência das perguntas, análise e<br/>interpretação dão voz aqueles que participaram.</li> </ul> |
| incluiu apenas um estudo quantitativo de Nível | <ul> <li>Interpretação perspicaz: Dados e conhecimentos estão ligados de maneira significativa à literatura relevante.</li> </ul> |
| III.<br>Estudos de meta-síntese -qualitativo. | C <u>Baixa qualidade</u> : Estudos de baixa qualidade contribuem pouco para, revisão geral dos resultados e tem pouco, se algum, dos recursos listados para alta / boa qualidade. |

Classificações de Qualidade

## Apêndice D

Nível de Evidencia e Guia de Qualidade

| Níveis de Evidência | Classificações de Qualidade |
|---|---|
| Nível IV Opinião de autoridades respeitadas e/ou de comitês formados por profissionais reconhecidos nacionalmente ou painéis de consensos baseados em evidências científicas. Incluindo: Diretrizes de prática clínica Painel de Consenso / Declarações de posicionamento | A <u>Alta Qualidade</u> : Meterial patrocinado oficialmente por organização profissional, pública ou privada, ou agência governamental; documentação de estratégia de pesquisa sistemática da literatura; resultados consistentes com números suficientes de estudos bem desenhados; avaliação baseada em critérios de força científica global e qualidade dos estudos selecionados; conclusões definitivas; conhecimento nacional evidente; desenvolvido ou revisado nos útimos 5 anos. B <u>Boa Qualidade;</u> ,,,,,Material patrocinado oficialmente por organização profissional, pública ou privada, ou agência governamental; documentação de estratégia de pesquisa sistemática da literatura adequada; resultados razoavelmente consistentes com números suficientes de estudos bem desenhados; avaliação de pontos fortes e limitações dos estudos selecionados; conclusões bastante definitivas, conhecimentos nacionais claramente evidentes; desenvolvido ou revisado nos últimos 5 anos. C <u>Baixa qualidade ou grandes falhas;</u> Material não patrocinado por uma organização ou agência oficial; estratégia de pesquisa da literatura indefinida, mal definida ou limitada; nenhuma avaliação dos pontos fortes e limitações dos estudos selecionados, evidências insuficientes com resultados inconsistentes, conclusões não podem ser definidas; não revisado nos últimos 5 anos. |
| Nível V Baseado em experiência e não evidencia de pesquisa. Inclui: Rexisões integrativas Rexisões de literatura Programas de melhoria de qualidade ou avaliação financeira Relatos de casos Opinião de especialista reconhecido nacionalmente baseado em evidência experimental | Experiência Organizacional (programas de melhoria de qualidade ou avaliação financeira) A Alta Qualidade: Objetivos claros; resultados consistentes em múltiplas configurações; métodos de avaliação de qualidade, financeiros, ou programas de melhoria (grapal, utilizados; conclusões definitivas; recomendações consistentes com referência aprofundada da evidência científica. B Boa Qualidade: Objetivos claros; resultados consistentes em uma única configuração; métodos de avaliação de qualidade, financeiros, ou programas de melhoria (grapal, utilizados; recomendações rezoavelmente coerentes com alguma referência de evidência científica. C Baixa qualidade ou grandes falhas: Objetivos não claros ou faltantes; resultados inconsistentes; melhoria de qualidade, financeiros, ou programas de avaliação de métodos mal definidos; recomendações não podem ser feitas. Revisão Integrativa, Revisão da Literatura, Opinião de Especialista, Relato de Casos, Padrão da Comunidade, Experiência Clínica, Preferência do Consumidor. A Alta Qualidade: A experiência é —evidente; delineia conclusões definitivas; fornece fundamentação científica; líder (es) de pensamento no campo ou área. B Boa Qualidade: A experiência aparenta ser credivel; tira conclusões bastante definitivas; fornece argumento lógico para opinões. C Baixa qualidade ou grandes falhas: A experiência não é discernível ou é duvidosa; conclusões não podem ser delineadas. |

1 https://www.york.ac.uk/erd/bysRev/ISSU/Webme.lp/E\_A\_ASSESSMENT\_OF\_Q.UAUTATIVE\_RESEARCH.htm 2 Adopted from Polit & Beak (2017).

## Apêndice E - Ferramenta de Avaliação de Evidência de Pesquisa

| Nível de evidência e classificação de qualidade: | |
|---|---|
| Título do artigo: | Número: |
| Autor (es): | Data de publicação: |
| Revista / Períodico: | |
| Configuração: | Amostra (composição e tamanho): |
| Essa evidência aborda minha pergunta de PBE? □ Sim □ Não – Não prossiga com a avaliação des | sa evidência |
| Este estudo é: | |
| Quantitativo (Coleta, análise e relato de dados numéricos). Dados mensuráveis (quantos; qual quantidade; ou quantas vezes) utilizados para formular fatos, descobrir padrões de pesquisa, e generalizar os resultados de uma amostra maior de população; fornece observação de efeitos de um programa, problema ou condição, medida com precisão, ao invés de interpretação dos dados pelo pesquisador. Métodos comuns são pesquisas, entrevistas face a face estruturadas, observações e revisões de registros ou documentos. Testes estatísticos são utilizados na análise dos dados. | |
| Ir para <u>Seção I: QuaNtitativo</u> | |
| Qualitativo (Coleta, análise e relato de dados narrativos). Documentos narrativos ricos são utilizados para descobrir temas; descrever problema ou condição do ponto de vista dos que experimentam. Os métodos comuns são grupos focais, entrevistas individuais (não estruturadas ou semi-estruturadas) e participação / observações. Tamanhos de amostras são pequenos e são determinados quando a saturação de dados é alcançada. A saturação de dados é atingida quando o pesquisador identifica que não surgem novos temas e a redundância está ocorrendo. A síntese é utilizada na análise dos dados. Frequentemente é um ponto de partida para estudos com pouca pesquisa existente; pode utilizar os resultados para projetar estudos empíricos. O pesquisador descreve, analisa e interpreta relatórios, descrições e observações dos participantes. | |
| Ir para <u>Seção II: QuaLitativo</u> | |
| Métodos mistos (resultados relatados numericamente e narrativamente). Ambos os métodos quantitativo e qualitativo são utilizados em projeto de estudo. Usando ambas as abordagens, em combinação, fornecem uma melhor compreensão dos problemas de pesquisa do que usar qualquer abordagem sozinha. Os tamanhos de amostras variam com base nos métodos utilizados. A coleta de dados envolve coletar e analisar dados quantitativos e qualitativos em único estudo ou série de estudos. A interpretação é continua e pode influenciar estágios no processo de pesquisa. | |
| Ir para <u>Seção I</u> para componentes <u>QuaNtitativos</u> e <u>Seção II</u> para componentes <u>QuaLitativos</u> | |

| Seção I: QuaNtitativo | | |
|---|---|---|
| Nível de Evidência (Desenho do Estudo) | | |
| A Isto é um relatório de um único estudo de pesquisa? | □ Sim | □Não<br><b>Ir para B</b> |
| 1. Houve manipulação de uma variável independente? | □ Sim | □ Não |
| 2. Havia um grupo controle? | □ Sim | □ Não |
| 3. Os participantes foram randomizados aos grupos de intervenção e controle? | □ Sim | □ Não |
| Se <b>Sim para as questões 1, 2, e 3,</b> este é um estudo experimental controlado randomizado (RCT) ou estudo experimental. | | NÍVEL I |
| Se Sim para questões 1 e 2 e Não para questão 3 ou Sim para questão 1 e Não para questões 2 e 3, este é quase-experimental. (Algum grau de controle do investigador, alguma manipulação de uma variável independente, falta de randomização aos grupos, e pode ter um grupo controle). | | NÍVEL II |
| Se Não para questões 1, 2, e 3, este é <u>não-experimental.</u> (Nenhuma manipulação de variável independente; pode ser descritivo, comparativo ou correlacional; frequentemente usa dados secundários). | | NÍVEL III |
| Achados do Estudo que ajudam a responder a pergunta de PBE: | | |
| Complete a Avaliação da seção de Estudos QuaNtitativos de Pesqu | isa | |

| Isto é um resumo de várias fontes de evidências de pesquisa? | □ Sim Continue | □ Não<br><b>Use Apêndice F</b> |
|---|---|---|
| Será que emprega uma estratégia de pesquisa abrangente e método de avaliação rigorosa? Se este estudo inclui pesquisa, não pesquisa, e evidências experienciais, é uma revisão integrativa (ver Apêndice F). | □ Sim<br>Continue | □ Não<br>Use Apêndice F |
| 2. Para revisões sistemáticas e revisões sistemáticas com meta-an | álise (veja as d | escrições abaixo): |
| a. Todos os estudos incluídos são RCTs? | | NÍVEL I |
| b. Os estudos são uma combinação de RCTs e quase-experimental? | ental, ou | NÍVEL II |
| c. Os estudos são uma combinação de RCTs, quase-experimental experimental, ou não experimental somente? | ntal, e não- | NÍVEL III |
| Uma revisão sistemática emprega estratégia de busca e método gera um tamanho de efeito. Uma meta-análise, ou revisão sistemática com meta-análise, com estudos para gerar uma nova estatística: o tamanho de efeito. Achados do Estudo que ajudam a responder a pergunta de PBE: | , | |
| Complete Avaliação da seção de Revisão Sistemática (com ou sem uma meta-análise) | | |

| Avaliação dos estudos de pesquisa QuaNtitativa | | | |
|---|---|---|---|
| O pesquisador identifica o que é conhecido e o que não é conhecido sobre o problema e como o estudo irá abordar quaisquer lacunas no conhecimento? | □ Sim | □ Não | |
| O objetivo do estudo foi claramente apresentado? | □ Sim | □ Não | |
| A revisão da literatura foi atual? (a maioria das fontes dentro dos últimos 5 anos ou um estudo seminal)? | □ Sim | □ Não | |
| O tamanho da amostra foi suficiente com base no projeto de estudo e racional? | □ Sim | □ Não | |
| Se houver um grupo controle: • As características e/ou demografia são similares nos grupos de controle e de intervenção? | □ Sim | □ Não | N/A |
| <ul> <li>Se múltiplas configurações foram utilizadas, foram configurações semelhantes?</li> </ul> | □ Sim | □ Não | N/A |
| <ul> <li>Todos os grupos foram tratados igualmente com<br/>exceção do (s) grupo (s) de intervenção?</li> </ul> | □ Sim | □ Não | N/A |
| Os métodos de coleta de dados são descritos claramente? | □ Sim | □ Não | |
| Os instrumentos foram confiáveis? (Alpha de Cronbach > 0.70)? | □ Sim | □ Não | N/A |
| A validade do instrumento foi discutida? | □ Sim | □ Não | N/A |
| Se foram utilizados <i>surveys</i> / questionários, a taxa de resposta foi > que 25%? | □ Sim | □ Não | N/A |
| Os resultados foram apresentados claramente? | □ Sim | □ Não | |
| Se tabelas foram apresentadas, a narrativa foi consistente com o conteúdo da tabela? | □ Sim | □ Não | N/A |
| As limitações do estudo foram identificadas e abordadas? | □ Sim | □ Não | |
| As conclusões foram baseadas nos resultados? | □ Sim | □ Não | |
| Ir para seção de Classificação de qualidade de estudos QuaNtit | ativos | | |

| Avaliação de Revisão Sistemática (com ou sem uma meta-análise) | | |
|---|---|---|
| As variáveis de interesse foram claramente identificadas? | □ Sim | □ Não |
| A pesquisa foi abrangente e reproduzível? • Principais termos de pesquisa indicados | □ Sim | □ Não |
| Múltiplos bancos de dados pesquisados e identificados | □ Sim | □ Não |
| Critérios de inclusão e exclusão indicados | □ Sim | □ Não |
| Houve um diagrama de fluxo que incluía o número de estudos eliminados em cada nível de revisão? | □ Sim | □ Não |
| Os estudos incluídos apresentados foram detalhados (desenho, amostra, métodos, resultados, desfechos, pontos fortes, e limitações)? | □ Sim | □ Não |
| Os métodos para avaliar a força e evidência (nível e qualidade) foram descritos? | □ Sim | □ Não |
| As conclusões foram baseadas nos resultados? | □ Sim | □ Não |
| Os resultados foram interpretados | □ Sim | □ Não |
| <ul> <li>As conclusões fluíram logicamente da interpretação e questão da<br/>revisão sistemática.</li> </ul> | □ Sim | □ Não |
| A revisão sistemática incluiu uma seção de endereçamento de limitações e como eles foram abordados? | □ Sim | □ Não |
| Complete seção Classificação de Qualidade para Estudos QuaNtitativos | | |

## Classificação de Qualidade para Estudos QuaNtitativos

Circule abaixo a classificação de qualidade apropriada:

- A Alta qualidade: Resultados consistentes e generalizados; tamanho de amostra suficiente para o desenho do estudo; controle adequado; conclusões definitivas; recomendações consistentes baseadas na revisão abrangente da literatura que inclui uma referência completa à evidência científica.
- **B** Boa qualidade: Resultados razoavelmente consistentes; tamanho de amostra suficiente para o desenho do estudo; algum controle, e conclusões bastante definitivas; recomendações razoavelmente consistentes baseadas em revisão de literatura bastante abrangente que inclui alguma referência à evidências científicas.
- **C** Baixa qualidade ou grandes falhas: Pouca evidência com resultados inconsistentes; tamanho de amostra insuficiente para o projeto de estudo; as conclusões não podem ser delineadas.

| Seção II: QuaLitativo | | |
|---|---|---|
| Nível de Evidência (Desenho do Estudo) | | |
| A lsto é um relatório de um único estudo de pesquisa? | □ Sim<br>Ir para Nível III | □ Não<br>Ir para II B |
| Achados do Estudo que ajudam a responder à pergunta de PBE: | | |
| Seção de Avaliação Completa de Estudo Único de Pesquisa QuaLitativa | | |

| Avaliação de um Estudo Único de Pesquisa QuaLitativa | | |
|---|---|---|
| Havia claramente identificável e articulado: • Objetivo? | □ Sim | □ Não |
| Pergunta de pesquisa? | □ Sim | □Não |
| Justificativa para método (s) utilizado (s)? | □ Sim | □ Não |
| Fenômeno que é o foco da pesquisa? | □ Sim | □ Não |
| A amostra de participantes foi representativa? | □ Sim | □Não |
| Possuem conhecimento ou experiência com a área da pesquisa? | □ Sim | □Não |
| As características dos participantes foram descritas? | □ Sim | □Não |
| A amostragem foi adequada, como evidenciado pela obtenção de saturação de dados? | □ Sim | □ Não |
| Análise dos Dados: | | |
| <ul> <li>Foi utilizado um processo de verificação a cada passo, verificando e<br/>confirmando com os participantes a confiabilidade da análise e<br/>interpretação?</li> </ul> | □ Sim | □Não |
| <ul> <li>Havia uma descrição de como os dados foram analisados (isto é,<br/>método), pelo computador ou manualmente?</li> </ul> | □Sim | □Não |
| Os achados suportam os dados narrativos (citações)? | □ Sim | □Não |
| Os achados fluem da pergunta da pesquisa aos dados coletados para a análise efetuada? | □ Sim | □Não |
| As conclusões são claramente explicadas? | □ Sim | □ Não |
| Ir para seção Classificação de Qualidade para Estudos QuaLitativos | | |

| В | Para resumos de múltiplos estudos de pesquisas qualitativas (meta-síntese) utilizou-se estratégia de pesquisa abrangente e um método de avaliação rigorosa? | □ Sim<br><b>Nível III</b> | □ Não<br>Ir para <b>Apêndice F</b> |
|---|---|---|---|
| Acha | ados do Estudo que ajudam a responder à pergunta de PBE: | | |
| Со | mplete a seção de Avaliação dos Estudos de Meta-Síntese | | |

| Avaliação dos Estudos de Meta-Síntese | | |
|---|---|---|
| A estratégia de busca e os critérios para a seleção de estudos primários foram claramente definidos? | □ Sim | □Não |
| Os achados foram apropriados e convincentes? | □ Sim | □ Não |
| A descrição dos métodos foram usadas para: • Comparar os resultados de cada estudo? | □ Sim | □Não |
| Interpretar dados? | □ Sim | □ Não |
| A síntese refletiu: | □ Sim | □ Não |
| Novas idéias? | □ Sim | □ Não |
| Descoberta de características essenciais dos fenômenos? | □ Sim | □ Não |
| <ul> <li>Uma compreensão mais completa dos fenômenos?</li> </ul> | □ Sim | □ Não |
| Os dados apresentados foram suficientes para apoiar as interpretações? | □ Sim | □ Não |
| Complete seção Classificação de Qualidade para Estudos QuaLitativos | | |

## Classificação de Qualidade para Estudos QuaLitativos

Circule abaixo a classificação de qualidade apropriada:

Não existem princípios comumente acordados para julgar a qualidade dos estudos qualitativos. É um processo subjetivo baseado na extensão em que os dados do estudo contribuem para a síntese e quanta informação é conhecida sobre os esforços dos pesquisadores para atender aos critérios de avaliação.

Para meta-sínteses, há concordância preliminar de que avaliações de qualidade individual dos estudos devem ser feitas antes da síntese para excluir estudos de baixa qualidade<sup>1</sup>.

A/B <u>Alta/Boa qualidade</u> é utilizada para estudos únicos e meta-sínteses<sup>2</sup>.

O relatório discute os esforços para melhorar ou avaliar a qualidade e a investigação geral com detalhes suficientes, descreve as técnicas específicas usadas para melhorar a qualidade da pesquisa.

Evidência de alguns ou todos os itens a seguir são encontrados no relatório:

- Transparência: Descrevem como as informações foram documentadas para justificar decisões, como os dados foram revisados por outras pessoas e como os temas e categorias foram formuladas.
- **Diligência:** Lê e reler os dados para checar interpretações, busca oportunidades para buscar múltiplas fontes para corroborar evidencias.
- Verificação: O processo de verificação, confirmação, e garantia de coerência metodológica.
- Auto-reflexão e escrutínio: Estar continuamente consciente de como as experiências, antecedentes ou preconceitos de um pesquisador pode moldar e influenciar análises e interpretações.
- **Pesquisa orientada por participantes:** Os participantes moldam o escopo e a abrangência das perguntas, análise e interpretação dão voz aqueles que participaram.
- **Interpretação perspicaz:** Dados e conhecimentos estão ligados de maneira significativa à literatura relevante.
- **C** <u>Baixa qualidade:</u> Estudos de baixa qualidade contribuem pouco para a revisão geral dos resultados e tem pouco, se algum, dos recursos listados c alta / boa qualidade.

## Seção III: Método Misto

## Nível de Evidência (Desenho do Estudo)

Você precisará avaliar de forma independente as partes quaNtitativas e quaLitativas do estudo, antes de avaliar o estudo em sua totalidade.

| a. Avalie a parte quaNtitativa do estudo usando a <b>Seção I.</b> | Nível | Qualidade |
|---|---|---|
| Insira aqui o nível de evidência e qualidade geral para esta parte. | | |

| b. Avalie a parte quaLitativa do estudo usando a <b>Seção II.</b> | Nív | el Q | ualidade |
|---|---|---|---|
| Insira aqui o nível de evidência e qualidade geral para esta parte. | | | |
| c. Para determinar o nível de evidência, circule o desenho de estudo apropriado | <b>)</b> : | | |
| <ul> <li>Explanatório sequenciais recolhem dados quaNtitativos primeiro, seguidos dos<br/>objetivo é explicar os resultados quaNtitativos usando os resultados quaLitativos<br/>baseado no nível da parte quaNtitativa.</li> </ul> | | | |
| <ul> <li>Exploratório sequenciais coletam dados quaLitativos primeiro, seguido dos dad<br/>objetivo é explicar os resultados quaLitativos usando os resultados quaNtitativos<br/>com base no nível da parte quaLitativa, e é sempre nível III.</li> </ul> | • | | |
| <ul> <li>Convergentes desenhos paralelos coletam os dados quaLititativos e quaNtitativos a finalidade de fornecer uma compreensão mais completa de um fenômeno, me de dados. Estes projetos são nível III.</li> </ul> | | | |
| <ul> <li>Multifásico coletam dados quaLitativos e quaNtitativos em mais de uma fase, c<br/>a próxima fase. Estes projetos são nível III.</li> </ul> | om cada | a fase in | formando |
| Achados do Estudo que ajudam a responder à pergunta de PBE: | | | |
| Use a seção de Avaliação de Estudos de Métodos Mistos | | | |
| Avaliação dos estudos de métodos mistos <sup>3</sup> | | | |
| O desenho da pesquisa de métodos mistos foi relevante para abordar as questões de pesquisa quaNtitativa e quaLitativa (ou objetivos)? | □ Sim | □ Não | □ N/A |
| O desenho da pesquisa foi relevante para abordar os aspectos quaNtitativos e quaLitativos da pergunta de métodos mistos (ou objetivos)? | □ Sim | □ Não | □ N/A |

pesquisa ou objetivos?

Para projetos paralelos convergentes, a integração dos dados quaNtitativos e quaLitativos (ou resultados) foram relevantes para abordar a pergunta da

□ Não

□ N/A

 $\square$  Sim

| Para projetos paralelos convergentes, as limitações associadas à integração (por exemplo, a divergência de dados quaLitativos e quaNtitativos ou resultados) foram suficientemente tratados? | □ Sim | □ Não | □ N/A |
|---|---|---|---|
| Ir para seção Classificação de Qualidade para Estudos de Métodos-Mistos | | | |

| Avaliação de Estudos Meta-Sínteses | | |
|---|---|---|
| As estratégias de busca e os critérios para seleção dos estudos primários foram claramente definidos? | □Sim | □Não |
| Os achados foram apropriados e convincentes? | □ Sim | □ Não |
| A descrição dos métodos utilizados foi: Comparar os resultados de cada estudo? | □ Sim | □Não |
| Interpretar dados? | □ Sim | □ Não |
| A síntese refletiu: | □ Sim | □ Não |
| Novas idéias? | □ Sim | □ Não |
| <ul> <li>Descoberta de características essenciais dos fenômenos?</li> </ul> | □ Sim | □ Não |
| <ul> <li>Uma compreensão mais completa dos fenômenos?</li> </ul> | □ Sim | □ Não |
| Os dados apresentados foram suficientes para apoiar as interpretações? | □ Sim | □ Não |
| Complete a seção de classificação de Qualidade de Estudos QuaLitativos | | |

3 National Collaborating Centre for Methods and Tools. (2015). Appraising Qualitative, Quantitative, and Mixed Methods Studies included in Mixed Studies Reviews: The MMAT. Hamilton, ON: McMaster University. (Updated 20 July, 2015) Retrieved from http://www.nccmt.ca/resources/search/232

## Classificação de Qualidade para Estudos de Métodos-Mistos

Circule a classificação de qualidade apropriada abaixo

- A <u>Alta Qualidade</u>: Contém componentes de estudos quaNtitativos e quaLitativos de alta qualidade; projeto de estudo altamente relevante; integração relevante de dados ou resultados; consideração cuidadosa das limitações da abordagem escolhida.
- **B** <u>Boa Qualidade:</u> Contém componentes de estudos quaNtitativos e quaLitativos de boa qualidade; projeto de estudo relevante; integração moderadamente relevante dos dados ou resultados; algumas discussões sobre as limitações da integração.
- C <u>Baixa qualidade ou grandes falhas:</u> Contém componentes de estudos quaNtitativos e qualitativos de baixa qualidade; projeto de estudo não é relevante para as questões da pesquisa ou objetivos; dados ou resultados mal integrados; nenhuma consideração dos limites de integração.

## <u>Apêndice F - Ferramenta de Avaliação de Evidências que não sejam de Pesquisa</u>

| Nível de Evidência e Classificação de Qualidade: | | | |
|---|---|---|---|
| Título do Artigo: | Número: | | |
| Autor(es): | Data de Publica | ação: | |
| Revista / Periódico: | | | |
| Configuração: | Amostra (comp | posição e tama | anho): |
| A evidência aborda minha pergunta de PBE? Sim Não- Não prossiga com a avaliação desta evidência | | | |
| □ Diretrizes de Prática Clínica - NÍVEL IV Recomendações sistematicamente desenvolvidas por especialistas reconhecidos nacionalmente com base em evidências de pesquisa ou painel de consenso de especialistas | | | |
| □ Consenso ou Declaração de Posição - NÍVEL IV Recomendações sistematicamente desenvolvidas, base especialistas reconhecidos nacionalmente, que orientam profissional na tomada de decisões para uma questão preoc | n os membros | | |
| Os tipos de evidências inclusos estão identificados? | | □ Sim | □ Não |

| <ul> <li>As partes interessadas (stakeholders) se envolveram no<br/>desenvolvimento de recomendações?</li> </ul> | □ Sim | □ Não |
|---|---|---|
| <ul> <li>As recomendações dos grupos aplicam-se e não se aplicam de forma<br/>clara?</li> </ul> | □ Sim | □ Não |
| Os possíveis vieses foram eliminados? | □ Sim | □ Não |
| Cada recomendação tem nível de evidência identificado? | □ Sim | □ Não |
| As recomendações são claras? | □ Sim | □ Não |
| Achados que ajudam a responder à pergunta de PBE: | | |
| Preencha a seção de classificação de qualidade correspondente | | |
| <ul> <li>Revisão de Literatura NÍVEL V Resumo da literatura publicada selecionada, incluindo científica e não cient experiência organizacional e opiniões de especialistas </li> <li>Revisão Integrativa NÍVEL V Resumo das evidências de pesquisa e literatura teórica; analisa, compara t literatura selecionada </li> </ul> | | |
| O assunto deve ser revisado claramente? | □ Sim | □ Não |
| <ul> <li>A literatura é relevante e atualizada (a maioria das fontes está nos últimos<br/>cinco anos ou clássica)?</li> </ul> | □ Sim | □ Não |
| <ul> <li>Da literatura revisada, há uma análise significativa das conclusões nos<br/>artigos incluídos na revisão?</li> </ul> | □ Sim | □ Não |
| Há lacunas identificadas na literatura? | □ Sim | □ Não |
| <ul> <li>As recomendações são feitas para a prática futura ou para o estudo?</li> </ul> | □ Sim | □ Não |
| Achados que ajudam a responder à pergunta de PBE: | | |
| Preencha a seção de classificação de qualidade correspondente. | | |

| <ul> <li>Opiniões de especialistas - NIVEL V</li> <li>Opinião de um ou mais indivíduos com base em experiência clí</li> </ul> | nica | | |
|---|---|---|---|
| O indivíduo publicou ou apresentou sobre o tópico? | | Sim | □ Não |
| A opinião do autor é baseada em evidências científicas? | | Sim | □ Não |
| A opinião do autor é claramente expressa? | | Sim | □ Não |
| Os possíveis vieses são reconhecidos? | | 3 Sim | □ Não |
| Achados que ajudam a responder à pergunta de PBE: | | | |
| Preencha a seção de classificação de qualidade corresponder | nte. | | |
| Experiência Organizacional | | | |
| <ul> <li>Melhoria da qualidade - NÍVEL V</li> <li>Método cíclico para examinar fluxos de trabalho, processos específica</li> <li>Avaliação financeira - NÍVEL V</li> <li>Avaliação econômica que aplica técnicas analíticas para identificant</li> </ul> | | | _ , |
| resultados de dois ou mais programas ou intervenções alternati Avaliação do programa - NÍVEL V Avaliação sistemática dos processos e/ou resultados de un quantitativos e qualitativos | vas | · | |
| Configuração: | Tamanho da | amostra/ ( | Composição: |
| O objetivo do projeto foi claramente identificado? | □ Sim | □ Não | ) |
| O método foi totalmente descrito? | □ Sim | □ Não | ) |
| As medidas de processo ou resultado foram identificadas? | □ Sim | □ Não | ) |
| Os resultados foram totalmente descritos? | □ Sim | □ Não | ) |
| A interpretação foi clara e apropriada? | □ Sim | □ Não | ) |
| <ul> <li>Os componentes da análise de custo/benefício ou custo-<br/>eficácia estão descritos?</li> </ul> | □ Sim | □ Não | o □ N/A |

| Achados que ajudam a responder à pergunta de | PBE: | | | | | |
|---|---|---|---|---|---|---|
| Preencha a seção de classificação de qua | lidade correspo | ndente. | | | | |
| □ Relato de caso - NÍVEL V Olhar aprofundado para pessoa, grupo ou | outra unidade soc | ial | | | | |
| ■ O objetivo do relato de caso é claramente | indicado? | | S | Sim | | Não |
| <ul> <li>O relato de caso está claramente apreser</li> </ul> | ntado? | | | Sim | | Não |
| As descobertas do relato de caso são apor<br>relevante? | oiadas por teoria o | u pesquisa | _ S | Sim | | Não |
| As recomendações estão claramente indi-<br>resultados? | cadas e estão ass | ociadas aos | _ S | Sim | | Não |
| Preencha a seção de classificação de qua | lidade correspo | ndente. | | | | |
| Padrão da comunidade, experiência do clír | nico ou preferên | cia do consi | umido | r - NÍVE | EL V | |
| Padrão da comunidade: Prática atual par | · | | | ade | | |
| □ Experiência do clínico: Conhecimento ao | • | | | . , | | |
| □ Preferência do consumidor: Conhecimer | nto adquirido atrav | es da experie<br>Número de f | | | | |
| Fontes de Informação (ões): | | inumero de f | onles. | | | |
| <ul> <li>Fonte de informação tem experiência<br/>credível</li> </ul> | □ Sim | □ Não | | | □ N/A | A |
| <ul> <li>As opiniões estão claramente<br/>indicadas</li> </ul> | □ Sim | □ Não | | | □ N/A | Α |
| <ul> <li>A evidência obtida é consistente</li> </ul> | □ Sim | □ Não | | | □ N/A | 4 |

| Achados que ajudam a responder à pergunta de PBE: |
|----------------------------------------------------------------|
| Preencha a secão de classificação de qualidade correspondente. |

Classificação de Qualidade para Diretrizes de Prática Clínica (*Guidelines*), Consenso ou Declarações de Posição (**Nível IV**)

#### A Alta Qualidade

Material oficialmente patrocinado por uma organização profissional, pública ou privada ou por uma agência governamental; documentação de uma estratégia sistemática de uma pesquisa bibliográfica; resultados consistentes com um número suficiente de estudos bem desenhados; avaliação baseada em critérios de força científica geral e qualidade dos estudos incluídos e conclusões definitivas; perícia nacional claramente evidente; desenvolvidos ou revisados nos últimos cincos anos.

## **B** Boa Qualidade

Material oficialmente patrocinado por organização profissional, pública ou privada ou por uma agência governamental; estratégia de busca sistemática de literatura razoavelmente completa e apropriada; resultados razoavelmente consistentes, número suficiente de estudos bem desenhados; avaliação das forças e limitações dos estudos incluídos com conclusões bastante definitivas; perícia nacional claramente evidente; desenvolvidos ou revisados nos últimos cinco anos.

#### C Baixa Qualidade ou Grandes Falhas

Material não patrocinado por organização ou agência oficial; estratégia de busca da literatura indefinida, mal definida ou limitada; nenhuma avaliação das forças e limitações dos estudos incluídos; evidência insuficiente com resultados inconsistentes; conclusões não podem ser delinadas; não revisado nos últimos cinco anos.

Classificação de Qualidade para Experiência Organizacional (Nível V)

## A Alta Qualidade

Objetivos e metas claras; resultados consistentes em várias configurações; melhoria formal da qualidade ou métodos utilizados de avaliação financeira; conclusões definitivas; recomendações consistentes com referência completa à evidências científicas.

#### **B** Boa Qualidade

Objetivos e metas claras; melhoria formal da qualidade ou métodos utilizados de avaliação financeira; resultados consistentes em uma única configuração; recomendações razoavelmente consistentes com alguma referência e evidências científicas.

## C Baixa Qualidade ou Grandes Falhas

Objetivos e metas pouca claras ou ausentes; resultados inconsistentes; qualidade mal definida; melhoria/ métodos de análise financeira; recomendações não podem ser feitas.

Classificação de Qualidade para Relato de Caso; Revisão Integrativa, Revisão da Literatura, Opinião de Especialista, Padrão da Comunidade, Experiência Clínica, Preferência do Consumidor (Nível V)

## A Alta Qualidade

O domínio é claramente evidente, tira conclusões definitivas e fornece uma justificativa científica; torna-se líder na área.

## **B** Boa Qualidade

O domínio parece ter credibilidade, delineia conclusões bastante definitivas e fornece opiniões e argumentos lógicos.

## C Baixa Qualidade ou Grandes Falhas

O domínio não é discernível ou é duvidoso; conclusões não podem ser delineadas.

## Apêndice G - Ferramenta de Evidência Individual

Apêndice G Ferramenta resumida de Evidência Individual

| Data: | | Questão PBE: | | | | | |
|---|---|---|---|---|---|---|---|
| Artigo.<br>Número. | Autor e Data | Jipo de<br>Exidência | Amostra,<br>Tamanho da<br>Amostra, Local<br>da Amostra. | Achados que ajudam a<br>responder a questão<br>de PBE | Medidas<br>observáveis | Limitações | Nível de Evidência.<br>Qualidade |
| | | | □ N/A | | | | |
| | | | □ N/A | | | | |
| | | | □ N/A | | | | |
| | | | D N/A | | | | |
| | | | □ N/A | | | | |
| | | | □ N/A | | | | |
| | | | □ N/A | etinos revisados o ara i | | | |

Anexe uma lista de referências com citações completas de artigos revisados para esta questão PEE

## Instruções para utilizar a Ferramenta resumida de Evidência Individual

## **Propósito**

Este formulário é utilizado para documentar os resultados da avaliação de evidências em preparação para a síntese de evidências.

O formulário fornece à equipe de PBE a documentação das fontes de evidências utilizadas, o ano que a evidência foi publicada ou de outra forma comunicada, a informação coletada de cada fonte de evidência que ajuda a responder à questão de PBE, e o nível e qualidade de cada fonte de evidência.

## **Artigo Número**

Atribua um número a cada fonte de evidência revisada. Isto organiza o resumo individual da evidência e possibilita uma maneira fácil de referenciar os artigos.

#### **Autor e Data**

Indique o sobrenome do primeiro autor ou a fonte de evidência e a data publicação/comunicação. Liste ambos autor/evidência e a data.

## Tipo de Evidência

Indique o tipo de evidência revisada (e.g., RCT, meta-análise, métodos mistos, qualitativo, revisão sistemática, estudo de caso, revisão narrativa de literatura).

## Amostra, Tamanho da Amostra, e Localização

Forneça uma rápida visualização da população, número de participantes, e local do estudo.

## Achados que ajudam a responder a questão de PBE

Embora, o revisor possa encontrar muitos pontos de interesse, liste apenas achados que aplicam diretamente para questão PBE.

## Medidas observáveis

Medidas quantitativas ou varáveis que são utilizadas para responder a pergunta de pesquisa, teste de hipóteses, descrever características, ou determinar o efeito, impacto ou influência. Evidência qualitativa utiliza casos, contextos, opiniões, experiências, e reflexões para representar o fenômeno do estudo.

## Limitações

Inclui informação que pode ou não estar dentro do texto do artigo sobre as desvantagens de uma parte da evidência. A evidência pode listar limitações, ou isto pode evidenciar para você, como rever a evidência, que um importante ponto é perdido ou a amostra não se aplica para a população de interesse.

#### Nível de Evidência e Qualidade

Utilize informação de ferramentas de avaliações individuais, transfira o nível de evidência e a classificação de qualidade para esta coluna.

## Apêndice H - Ferramenta de Síntese de Evidências e Recomendações

## Apêndice H

Ferramentas de Sínteses de Processos e Recomendações



#### **Pontos-Chaves:**

Síntese de Evidência é o melhor executada por meio da discussão em grupo.
Todos os membros da equipe dividem suas perspectivas, e a equipe utiliza o
pensamento crítico para chegar a um julgamento consensuado durante o
processo de síntese. O processo de síntese envolve tanto razões subjetivas
quanto objetivas de raciocínio de toda a equipe de PBE.

Por meio do raciocínio, a equipe:

- Revisar a avaliação da qualidade de peças individuais de evidência
- Avalia e assimila consistências nos resultados
- Avalia o significado e a relevância dos resultados
- Mescla resultados que podem aprimorar o conhecimento da equipe ou gerar novos insights, perspectivas e entendimentos
- Destaca inconsistências nos resultados
- Faz recomendações com base no processo de síntese
- Quando a evidência inclui múltiplos estudos de evidência no Nível I e Nível II, há uma população semelhante ou definição de interesse, e há consistência por meio de resultados, o time de PBE pode ter maior confiança em recomendar uma mudança na prática. No entanto, com a maioria das evidências de Nível II e Nível III, a equipe deve proceder com cautela ao fazer mudanças na prática. Neste instante, as recomendações tipicamente incluem a conclusão de um piloto antes de decidir implementar uma mudança em grande escala.
- Geralmente, mudanças na prática não são feitas na evidência de Nível IV ou V.
   No entanto, as equipes têm uma variedade de opções para ações que incluem, mas não se limitam a: criação de campanhas de conscientização, realização de atualizações informativas e educacionais, monitoramento de fontes de evidência para novas informações e elaborações de estudos de pesquisa.
- A classificação de qualidade (veja Apêndice D) é para avaliar tanto evidências de qualidade individuais quanto gerais.
### Apêndice H

. Ferramentas de Sínteses de Processos e Recomendações

| Questão PBE: | | | |
|---|---|---|---|
| Categoria (Tipo de Nível) | Número Total de<br>Fontes/Nível | Classificação<br>Geral de<br>Qualidade | Síntese de Resultados<br>Evidência das Respostas da Questão PBE |
| Nível, I Studo experimental Tracio Jandounizado Controlado (ERC) Levisões Sistemálicas do EIC com ou sem meta-análise Desenho do método misto explora tório que inclui apenas um estudo qualitativo Hivel I | | | |
| Nível II Estudos quase-experimentais Revisão systemática da combinação de ERC e estudos quase-experimentais, ou apenas quase-experimentais, com ou sem meta-análise Desenho do método misto exploratório que inclui somente o estudo qualitativo Nível II | | | |
| Nível III Estudo não experimental Revisão sistemática da combinação de ERCs, estudos quaserexperimental e não experimental, ou apenas estudos não experimentais, com ou sem meta-análise Estudo qualitativo ou meta-síntese Exploratório, convergente ou métodos de estudos mistos e multifásicos. Desenho exploratório misto que inclui somente o estudo qualitativo Nível III | | | |

### Apêndice H

. Ferramentas de Sínteses de Processos e Recomendações

| Categoria (Tipo de Nível) | Número Total de<br>Fontes/Nível | Classificação<br>Geral de<br>Qualidade | Síntese de Resultados<br>Evidência das Respostas da Questão PBE |
|---|---|---|---|
| Nível IV Opiniões de autoridades respeitadas e/ou relatório de comitês de especialista reconhecidos nacionalmente ou painéis consensuais baseados na evidência científica | | | |
| Nível V • Evidência da lileratura ou revisão integrativa, melhoria de qualidade, avaliação do programa, avaliação financeira ou relatos de caso. | | | |
| <ul> <li>Opinião de especialistas reconhecidos<br/>nacionalmente baseados na evidência<br/>experimental.</li> </ul> | | | |

# Baseado em sua síntese, quais dos quatros caminhos a seguir traduzem a representação da força total da evidência? | Forte, evidência convincente, resultados consistentes: Indicação sólida para uma mudança de prática é indicada. | Evidência boa e consistente: Considere piloto de mudança ou investigação adicional. | Evidência boa, mas conflitante: Não indicado para mudança de prática; considere investigação adicional para nova evidência ou desenvolver um estudo de pesquisa. | Pouca ou nenhuma evidência: Não indicado para mudança de prática; considere investigação adicional para nova evidência, desenvolver estudo de pesquisa, ou descontinuação de projeto. Se você selecionou a primeira opção ou a segunda opção, continue. Do contrário, PARE, a tradução não é indicada. Recomendações baseadas na síntese de evidência e caminho de tradução selecionado

### Considere o seguinte ao examinar os ajustes:

As recomendações são:

- Compatível com a cultura, os valores ou normas da unidade / departamento / organização?
- Consistente com os assuntos, as estruturas, atitudes, crenças e/ou práticas da unidade / departamento / organização?
- Consistente com as prioridades da unidade/departamento/organização?

### Considere o seguinte ao examinar a viabilidade:

- Podemos fazer o que eles fizeram no nosso ambiente de trabalho?
- Os seguintes suportes estão disponíveis?
  - Recursos
  - Financiamento
  - Aprovação de líderes administrativos e clínicos
  - Suporte de partes interessadas
- É provável que as recomendações possam ser implementadas dentro da unidade / departamento / organização?

### Instruções para uso deste formulário:

### Objetivo do formulário

Utilize este formulário para compilar os resultados da avaliação individual de evidências para responder à pergunta da PBE. Os achados pertinentes para cada nível de evidência são sintetizadas, e uma classificação de qualidade é atribuída a cada nível.

### Número total de fontes por nível

Registre o número de fontes de evidência para cada nível.

### Classificação geral de qualidade

Resume a qualidade geral da evidência para cada nível. Utilize o Apêndice D para classificar a qualidade da evidência.

### Síntese de achados: evidência de respostas da pergunta PBE

- Inclua somente achados de qualidade de evidência A ou B.
- Inclua apenas declarações que respondem diretamente a questão PBE.
- Resuma os resultados/achados dentro de cada nível de evidência.
- Registro o(s) número(s) de artigo(s) do resumo de evidência individual entre parênteses ao lado de cada declaração para que a origem do resultado seja fácil de identificar.

# Desenvolver recomendações baseadas na síntese de evidência e o caminho da tradução selecionada

Revise os achados da síntese e determine quais dos quatro caminhos para tradução representam a força total da evidência:

- Forte, evidência convincente, resultados consistentes: Indicação sólida para mudança de prática.
- Evidência boa e consistente: Considere piloto de mudança ou investigação adicional.
- Evidência boa, mas conflitante: Não indicada para mudança de prática, considere investigação adicional para nova evidência ou desenvolvimento de pesquisa
- Pouca ou nenhuma evidência: Não indicado para mudança de prática; considere investigação adicional para nova evidência, desenvolver um estudo de pesquisa, ou descontinue o projeto.

### Ajuste e viabilidade

Mesmo quando a evidência é forte ou de alta qualidade, pode não ser apropriado implementar mudança na prática. É crucial examinar a viabilidade que considera os recursos disponíveis, a prontidão para a mudança e o equilíbrio entre o risco e o benefício. O ajuste refere-se à compatibilidade da mudança proposta com a missão, metas, objetivos e prioridades da organização. Uma mudança que não se enquadre nas prioridades organizacionais terá menos probabilidade de receber suporte da liderança e apoio financeiro, dificultando o sucesso. A implementação de processos com baixa probabilidade de sucesso desperdiça tempo e recursos valiosos em esforços que produzem benefícios negligenciáveis.

# Apêndice I - Ferramenta de Planejamento de Ações

| 1. Complete as seguintes atividades para garantir uma tradução bem sucedida: | | |
|---|---|---|
| □ Identifique um líder do projeto. | | |
| □ Identifique responsáveis pelas mudanças. | | |
| □ Considere incluir membros | ou diferentes atividades durante | e a tradução do projeto. |
| □ Agende tempo suficiente pa | ra completar as tarefas principa | ais. |
| □ Identifique tarefas cruciais e | atividades relacionadas. | |
| ☐ Identifique medidas pré ou p | oós observacionais. | |
| 2. Identifique barreiras para o sucesso da mudança, e então identifique forças que podem alavancar e superar barreiras | | |
| Barreiras | Pesquisas ou Forças | Planeje superar barreiras, aproveitando os pontos fortes como apropriado |
| 3. Considere ou como esta | mudança afetará o segui | nte: |
| | ☐ Registro eletrônico de sau | úde |
| Fluxo de trabalho | □ Política | as e/ou procedimentos |
| 4. Confirme o suporte e/o (Verifique todos que se | - | dos para cobrir as despesas. |
| □ Custos pessoais | s □ Educ | ☐ Educação ou aperfeiçoamento |
| □ Suprimentos/Eq | uipamentos 🖵 Cont | ☐ Conteúdo ou especialistas externos |
| □ Tecnologia | □ Cust | os da Disseminação (custos de viagem |
| □ Fotocópias | custo | os da conferência) |
| · | □ Outr | 0: |

| 5. Identificar pontos críticos e tarefas relacionadas: | | | | |
|---|---|---|---|---|
| | (Inserir ponto 1) | (Inserir ponto 2) | (Inserir ponto 3) | (Inserir ponto 4) |
| | (Inserir tarefa) | | | |
| S | | | | |
| Tarefas | | | | |

### Instruções para uso da ferramenta de planejamento de ações

### Objetivo do formulário

Este formulário é utilizado para guia-lo ao criar um plano de ação.

### Atividades para garantir uma tradução bem-sucedida

Essas são todas as atividades que devem ser concluídas à medida que você planeja a mudança. Considere as medidas pré e pós-observáveis que podem ser usadas para determinar se a mudança foi bem-sucedida. Além disso, a identificação de pontos críticos permite que a equipe veja se eles estão no caminho certo para atingir as metas.

# Identifique pontos fortes/ recursos e barreiras para o sucesso da mudanca

Análise que permite as equipes identificarem barreiras à implementação e, potencialmente reduzi-las por meio de forças e recursos inerentes. Pode-se encontrar desafios específicos que provavelmente afetarão a capacidade de cumprir o plano de ação. Embora esses obstáculos possam atrapalhar, o conhecimento deles é útil para que você possa envolver o suporte e criar um plano para resolvê-los.

# Considere se ou como a alteração afetará fluxos de trabalhos e processos

Esteja ciente do impacto da mudança. Por exemplo, será necessário fazer alterações no prontuário eletrônico para acomodar a alteração ou essa mudança afetará o fluxo de trabalho de qualquer outra equipe que tenha sido considerada?

### Confirme o apoio e/ou disponibilidade de fundos para cobrir despesas

Use isso como um guia para alertar sobre as obrigações financeiras que podem fazer parte do lançamento.

### Identificar pontos críticos e tarefas relacionadas

Considere todas as categorias de trabalho (pontos) necessários para implementar essa mudança. Quais tarefas devem ser realizadas em um primeiro momento para cada ponto a fim de avançar? Quando eles devem ser concluídos para permanecer no caminho certo? Por exemplo, se o ponto for implementar protocolo, listar todas as tarefas para realiza-lo.

# Apêndice J - Ferramenta de Disseminação

| 1. Pense sobre as descobertas do projeto e pratique a iniciativa de mudança. Qual é a informação mais importante que você precisa transmitir? | | |
|---|---|---|
| 2. Alinhar mensagens-chave | s com os públicos-alvo | |
| Público Alvo | Mensagem-chave | Método de Comunicação |
| Interdisciplinaridade das partes interessadas (stakeholders) | | |
| Liderança Organizacional | | |
| Liderança por Departamento | | |
| Equipe da Linha de Frente | | |
| Comunidade Externa<br>(publicações, pôsteres, e<br>apresentações) | | |
| 3. Análise dos exemplos ab apropriados | aixo para identificar os métodos | de comunicação |
| <ul> <li>Publicação Escrita</li> <li>Programa Online</li> <li>Conferência Externa</li> <li>Apresentação oral</li> <li>Apresentação de poster</li> <li>Publicação em mídia social</li> <li>Reunião interna/ no serviço</li> <li>Conteúdo de áudio/vídeo</li> <li>Outros:</li> </ul> | | |

### Instruções para uso da ferramenta de disseminação

### Objetivo

Esta forma é útil de vários pontos no processo do projeto PBE. Geralmente é concluída no final do projeto, quando os achados são conhecidos e os esforços produziram um produto, uma ferramenta, um programa ou uma política.

### Alinhar a mensagem chave com o público-alvo

Pense sobre os achados do projeto. Qual foi a conquista obtida com o projeto? Quais os produtos, as mudanças da política ou resultados que você pode relatar? Identificar os usuários finais – quem é seu público alvo? Seu público alvo pode ser individual, organizacional ou redes que possam ter interesse nos resultados do projeto.

### Método de comunicação

Este é o plano de comunicação e pode ocorrer em muitos níveis. Pense sobre alcançar diversos públicos utilizando uma infinidade de métodos. Estes podem estar inclusos, mas não é limitado para escrita, para o conteúdo visual/áudio, programas online e apresentações de pôster.

# Appendix 4:

STRUCTURING ASSESSMENT QUESTIONNAIRE AND DESCRIPTION OF A PRACTICE PROJECT BASED ON EVIDENCE FROM THE CLINICAL NURSE'S PERSPECTIVE

| Full na | ame: |
|---|---|
| | <del>-</del> |
| 1. | Think about the time to describe the clinical question based on the example of a problem, this was: |
| | ( ) very slow ( ) slow ( ) fast ( ) very fast |
| 2. | Looking for an evidence in the database was: |
| | ( ) challenging ( ) difficult ( ) easy ( ) very easy |
| 3. | In relation to critical analysis and quality classification, the |
| | understanding of scientific articles was: |
| | ( ) not understandable ( ) partially understandable |
| | ( ) understandable ( ) totally understandable |
| 4. | Summarize and classify the levels of evidence was: |
| | ( ) challenging ( ) difficult ( ) easy ( ) very easy |
| 5. | The description of the feasibility of applying the evidence was: |
| | () challenging () difficult () easy () very easy |
| 6. | The development of an action plan for the dissemination of |
| | evidence was: |
| | ( ) not helpful ( ) partially helpful ( ) helpful ( ) very helpful |
| 7. | In relation to going through the phases of an evidence-based |
| | practice project, the material offered during the workshop was: |
| | ( ) not helpful ( ) partially helpful ( ) helpful ( ) very helpful |

| B. Additional comments: |
|-------------------------|

# Appendix 5:

# COMPLIANCE VERIFICATION QUESTIONNAIRE IN THE EXERCISE OF PREPARING a PBE PROJECT, FROM THE RESEARCHER'S PERSPECTIVE

| Re | esearch | ner's r | name: | | | | | | _ |
|---|---|---|---|---|---|---|---|---|---|
| Pa | ırticipa | nt's na | ame: | | | | | | |
| ( | ) Gro | up A | ( | ) Gro | oup B | | | | |
| | 1. | Was | the par | ticipar | nt able to ela | bora | te a cli | nical question? | |
| | | | ( | ) Yes | 5 | | ( | ) No | |
| | 2. | The | survey | of bibl | iographic ar | ticles | s was | | |
| | ( ) Sufficient ( ) Partially sufficient ( ) Insufficient | | | | | | | | |
| | 3. | Reg | arding t | he clas | ssification o | f evic | dence a | according to the level o | f |
| | | qual | ity, was | the pa | articipant ab | le to | carry o | out this classification? | |
| | | ( | ) Yes | ( | ) Partially | ( | ) No | | |
| | 4. | Was | the par | ticipar | nt able to ela | bora | te a sy | nthesis of the findings | |
| | | relat | ing to tl | ne leve | els of eviden | ice? | | | |
| | | ( | ) Yes | ( | ) Partially | ( | ) No | | |
| | 5. | 5. W | as the p | articip | ant able to | devel | lop a d | issemination plan for | |
| | | impl | ementir | ng the | PBE project | ? | | | |
| | | ( | ) Yes | ( | ) Partially | ( | ) No | | |

### Appendix 6:

### **Program content:**

### Lesson Plan - THEORETICAL-PRACTICAL WORKSHOP

Model: Presencial Hours: 6 hours

Menu: The workshop proposes a review of all stages of EBP which includes approaches to clinical care based on science and the quality of evidence, with the ultimate goal of promoting safe and quality care.

### **Program content:**

Teaching strategies (methodologies): Lecture / Mini-lecture / Kahoot:

- Introduction to PBE
- Identification of a problem and elaboration of a clinical question
- Video lesson on searching for evidence and using a scientific database
- Classification of evidence levels / summary of evidence
- Elaboration of an action plan for the implementation of evidence-based clinical practice
- Dissemination and sharing of the project.

### Practical Lesson (case exercise):

### Case 1 group description:

Structuring a PBE project based on the knowledge acquired in the initial topics of the Workshop

To base this exercise, we will use a finalized and consolidated project, which will be used as a template for the exercise.

The participant will receive the description of a problem as a basis for elaborating their clinical question and thus go on to the following phases.

From that point on, the participant will be free to go through the following phases based on the previous content received the previous day, no sequence will be provided to follow the project.

To search for scientific evidence, access to a computer room will be offered to conduct research in the databases: PUBMED and CINAHL.

For the evaluation of evidence, we will not use articles from the results of each participant. 2 articles previously classified in the final PBE project will be delivered so that the participant can carry out their classification of level and quality of evidence of these articles. The form of classification of the participant will be compared with the previous classification and used to assess this requirement in the questionnaire to verify compliance in the exercise of preparing a PBE project from the researcher's perspective.

In continuation of the workshop and based on these 2 articles, the participant must prepare a summary of the findings relating to the levels of evidence found and recommendations.

The finalization will be with the elaboration of a plan for the dissemination of these results, which should involve the interested parties in the PBE project in question.

### **Group 2 case description:**

It will follow the same molds as the case of group 1 plus the Johns Hopkins Nursing Evidence-based Practice forms since the beginning of this practical class, when the participant will receive a description of a problem as a basis for elaborating their clinical question and thus go to the stage following.

The following forms will be offered in the case of this group: question development, evidence level and quality guide, research evidence assessment tool, individual evidence tool, evidence synthesis and recommendation tool, action planning tool and tool dissemination.